Statistical Analysis Plan

Study Code C2661002

Edition Number 2.7

Date 22 March 2018

Open-label, Multicentre Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ceftaroline in Neonates and Young Infants with Late-Onset Sepsis

Open-label, Multicentre Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ceftaroline in Neonates and Young Infants with Late-Onset Sepsis

#### Statistical Analysis Plan

Study Code

C2661002

Edition

2.7

Number

Date 22 March 2018

Open-label, Multicentre Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Ceftaroline in Neonates and Young Infants with Late-Onset Sepsis

# SIGNATURE OF GLOBAL PRODUCT STATISTICIAN



| TABLE | E OF CONTENTS | PAGE |
|---|---|---|
| TITLE PA | AGE | 1 |
| SIGNAT | URE OF STUDY STATISTICIAN | 2 |
| SIGNAT | URE OF GLOBAL PRODUCT STATISTICIAN | 3 |
| TABLE ( | OF CONTENTS | 4 |
| LIST OF | ABBREVIATIONS | 6 |
| AMEND | MENT HISTORY | 8 |
| 1. | STUDY DETAILS | 11 |
| 1.1<br>1.1.1<br>1.1.2<br>1.1.3 | Study objectives Primary objective Secondary objectives Exploratory objectives (Not applicable) | 11 |
| 1.2 | Study design | 11 |
| 1.3 | Number of patients | 17 |
| 2. | ANALYSIS SETS | 17 |
| 2.1<br>2.1.1<br>2.1.2<br>2.1.3<br>2.1.4<br>2.1.5 | Definition of analysis sets Intent-to-treat Analysis Set Safety Analysis Set Modified Intent-to-Treat Analysis Set Microbiological Intent-to-Treat Analysis Set Pharmacokinetic (PK) Analysis Set | 17<br>18<br>18 |
| 2.2 | Protocol deviations. | 18 |
| 3. | PRIMARY AND SECONDARY VARIABLES | 18 |
| 3.1<br>3.1.1<br>3.1.1.1<br>3.1.1.2<br>3.1.1.3<br>3.1.1.4<br>3.1.1.5 | Primary outcome variables. Safety variables. Adverse events (AE) variables. Death Clinical laboratory variables Vital signs variables Other safety variables. | 19<br>20<br>20<br>21 |
| 3.2<br>3.2.1<br>3.2.1.1<br>3.2.1.2 | Secondary outcome variables Efficacy variables Clinical response variable at EOT and TOC Per-pathogen and per-patient microbiological response variables at EOT and TOC | 22 |
| 3.2.2<br>3.3.1<br>3.3.1.1 | Pharmacokinetic variables Demographic and baseline characteristic variables Demographic variables | 26<br>27 |

| 3.3.1.2 | Surgical and medical history variables including antepartum/ | 27 |
|---|---|---|
| 2 2 1 2 | peripartum period | 27 |
| 3.3.1.3 | Baseline microbiological assessment variables for blood, CSF, urine, | 27 |
| 2.2.2 | and other specimens | |
| 3.3.2 | Definition of prior and concomitant medication | |
| 3.3.3 | Exposure and Compliance variable | 28 |
| 4. | ANALYSIS METHODS | 29 |
| 4.1 | General principles | 29 |
| 4.1.1 | Data quality | 29 |
| 4.2 | Analysis methods | 29 |
| 4.2.1 | Patient disposition | 29 |
| 4.2.2 | Protocol deviations. | 30 |
| 4.2.3 | Demographics and baseline characteristics | 30 |
| 4.2.4 | Prior and concomitant medications. | |
| 4.2.5 | Study therapy exposure and compliance | 31 |
| 4.2.6 | Safety analysis | |
| 4.2.6.1 | Analysis of adverse events, serious adverse events, and deaths | |
| 4.2.6.2 | Clinical laboratory safety assessment | |
| 4.2.6.3 | Weight, vital signs, and oxygen saturation results | |
| 4.2.6.4 | Other safety results | |
| 4.2.7 | Efficacy analysis | |
| 4.2.7.1 | Clinical response | |
| 4.2.7.2 | Microbiological response | |
| 4.2.8 | Pharmacokinetics analysis | |
| 5. | APPENDICES | 33 |

# LIST OF ABBREVIATIONS

| Abbreviation or special term | Explanation |
|------------------------------|----------------------------------------------|
| AE | Adverse event |
| AESI | Adverse event of special interest |
| BE | Base excess |
| BLQ | Below limit of quantification |
| CBC | Complete blood count |
| CI | Confidence interval |
| CRF | Case report form |
| CRP | C-reactive protein |
| CSF | Cerebrospinal fluid |
| CT | Computed tomography |
| CTMS | Clinical Trials Management System |
| CV | Coefficient of variation |
| CXR | Chest radiograph |
| DSMB | Data Safety Monitoring Board |
| EOT | End-of-therapy |
| ICF | Informed consent form |
| ITT | Intent-to-treat |
| IV | Intravenous |
| LLN | Lower limit of normal |
| LOS | Late-onset sepsis |
| LOQ | Limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MIC | Minimum Inhibitory Concentration |
| MITT | Modified intent-to-treat |
| MRI | Magnetic resonance imaging |
| NC | Not calculable |
| NQ | Non quantifiable |
| OAE | Other significant AE |
| PCS | Potentially clinically significant |
| PD | Protocol deviation |
| PK | Pharmacokinetic |
| q8h | Every 8 hours |

| Abbreviation or special term | Explanation |
|---|---|
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SFU | Safety follow-up |
| SMQ | Standard MedDRA Query |
| SOC | System organ class |
| TFL | Tables, Figures and Listings |
| TOC | Test-of-cure |
| ULN | Upper limit of normal |
| WBC | White blood cell |
| WHODDE | World Health Organization Drug Dictionary Enhanced |

# **AMENDMENT HISTORY**

| Date | Brief description of change |
|---|---|
| 9 Dec 2014 | V0.1 |
| | Initial Statistical Analysis Plan (SAP) for client review. |
| 7 Jan 2015 | V0.2 |
| | Version incorporating client review comments on V0.1. |
| 21 Jan 2015 | V1.0 |
| | Signed version approved for programming commencement incorporating client review comments on V0.2. |
| 8 June 2016 | V2.0 |
| | Updated version of the SAP incorporating Protocol Amendment changes as outlined below: |
| | Change in definition of study day from "Study Day 1 is defined as the first day of study therapy administration." to "Study Day 1 will start at the onset of study therapy and will end 24 hours later.". Change in definition of cohort 2 from "Cohort 2: term neonates (defined as gestational age ≥38 weeks) aged 7 to ≤28 days". to "Cohort 2: term neonates (defined as gestational age ≥37 weeks) aged 7 to ≤28 days". Change in definition of cohort 3 from "Cohort 3: preterm neonates (defined as gestational age ≥34 to <38 weeks) aged 7 to ≤28 days" to "Cohort 3: preterm neonates (defined as gestational age ≥34 to <37 weeks) aged 7 to ≤28 days". Change in dose from "Ceftaroline fosamil will be given at a dose of 4 mg/kg IV over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour)." to "Ceftaroline fosamil will be given at a dose of 6 mg/kg IV over 60 (± 10) minutes every 8 hours (q8h) (± 1 hour).".]. Change in requirements for administration of IV ampicillin and optional aminoglycoside from "IV ampicillin and optional aminoglycoside will be given as per standard of care." to "IV ampicillin and optional aminoglycoside will be given as per standard of care. If the presence of an organism that requires treatment with ampicillin cannot be excluded, then the use of IV ampicillin for the first 48 hours is mandatory. If the result of additional microbiology, polymerase chain reaction or other investigations, indicate that ampicillin during the first 48 hours of treatment is not required, then its use is at the discretion of the investigator.". |
| | In addition to the changes in relation to protocol amendments, additional tables were added for the duration of different Investigational Products (IP) [Ceftaroline, Ampicillin and Aminoglycoside]. Some additional programming notes were added to the shells to assist with the definition of variables within the derived/analysis datasets. An additional appendix was added to the SAP to list the criteria for |
| | potentially clinically significant laboratory tests. An additional appendix was added to the SAP to indicate the TFLs required |

| Date | Brief description of change |
|---|---|
| 12 July 2016 | V2.1 |
| | Updated to incorporate client review comments on V2.0. |
| | Updated to incorporate protocol amendment 2 changes: study medication dose changed from 4mg/kg to 6mg/kg. |
| 23 August 2016 | V2.2 |
| | Updated to incorporate client review comments on V2.1: In section 3.1.1.1, if the intensity of an Adverse Event (AE) is missing, the AE will be regarded as having missing rather than severe intensity; If the relationship of an AE to IMP is missing, the AE will be regarded as having a missing relationship to IMP rather than being related to IMP; and |
| | an additional table for the duration of prior medication was added. |
| | Updated to incorporate protocol amendment 3 changes: inclusion criteria 3, 4 and 5 were revised so that patients must meet at least 1 of the listed laboratory criteria, rather than 2 of the criteria and justification provided for the dose increase to 6mg/kg in the previous protocol amendment. |
| 5 September 2016 | V2.3 |
| • | Additional details added to the amendment history for V2.2 of the SAP. |
| | The text of SAP Appendix A was clarified. |
| | Listing was replaced with Appendix in the "Source:" footnote of Tables. |
| | Listing xx.x.xx was removed from the footnotes of the TFL appendix shells, as not required. |
| 6 December 2017 | V2.4 |
| | Updated to incorporate protocol amendment 4. Version of protocol and CRF updated. Additional Tables and Listings added further to receipt of Pfizer review |
| | comments. |
| | Unnecessary appendices removed and cross-references within the SAP updated. |
| | Details in relation to the DSMB modified and DSMB Tables and Listings removed as no further DSMBs to occur. |
| 12 January 2018 | V2.5 |
| | Updated to incorporate final Pfizer review comments on V2.4 SAP and TFL shells. |
| | Additional Tables and Listings added. |
| | Further TFL numbering changes incorporated. |
| | Additional Microbiological ITT population added. |
| | Further clarification of non-eligible organisms provided in Appendix A. |
| 16 March 2018 | V2.6 |
| | Incorporate final changes to the SAP ahead of database lock. |
| | Update to include list of AESIs. |
| | Update to Micro-ITT population definition. |
| | Post Data Review Meeting changes incorporated. |

Date Brief description of change

22 March 2018 V2.7

Appendix A updated to move Enterococcus species from never to sometimes a pathogen based on investigator determination.

Statistical Analysis Plan Study Code C2661002 Edition Number 2.7 Date 22 March 2018

#### 1. STUDY DETAILS

This statistical analysis plan (SAP) describes the statistical methods to be used during the reporting and analyses of data collected under Pfizer Protocol C2661002. This version of the plan has been developed using the protocol dated 25 May 2017 and case report form (CRF) dated 17 November 2017. Any further changes to the protocol or CRF may necessitate updates to the SAP and will be captured in an amendment.

# 1.1 Study objectives

### 1.1.1 Primary objective

The primary objective is to evaluate the safety and tolerability of ceftaroline for the treatment of late-onset sepsis (LOS) in neonates and young infants aged 7 to <60 days.

#### 1.1.2 Secondary objectives

The secondary objectives are:

- To evaluate the pharmacokinetic (PK) profile of ceftaroline in neonates and young infants aged 7 to <60 days with LOS
- To evaluate the efficacy of ceftaroline for the treatment of LOS in neonates and young infants aged 7 to <60 days.

#### 1.1.3 Exploratory objectives (Not applicable)

## 1.2 Study design

This open label, multicentre, multinational, single treatment arm study will evaluate the safety, tolerability, PK, and efficacy of ceftaroline fosamil and ampicillin, plus an optional aminoglycoside of choice, in hospitalized neonates and young infants with LOS. The study will be conducted in approximately 30 centres worldwide. Eligible pediatric patients (7 to <60 days) with suspected or confirmed LOS will be enrolled in this study. At least 24 patients with LOS will be enrolled and treated within three age cohorts of 8 patients:

- Cohort 1: young infants aged >28 days to <60 days (n=8)
- Cohort 2: term neonates (defined as gestational age ≥37 weeks) aged 7 to ≤28 days (n=8)
- Cohort 3: preterm neonates (defined as gestational age ≥34 to <37 weeks) aged 7 to ≤28 days (n=8).

This study is not randomized, but patients will be stratified by age cohort and randomly assigned (1:1) at the time of enrolment to 1 of the PK sample collection schedules:

- PK Schedule 1: at the end of the ceftaroline fosamil infusion (± 5 minutes, i.e. within 5 minutes of the end of the ceftaroline infusion) and 3 to 4 hours after the end of the infusion
- PK Schedule 2: 15 minutes to 2 hours after the end of the ceftaroline fosamil infusion and 5 to 7 hours after the end of the infusion (before the start of the next infusion).

Study therapy will consist of standard of care ampicillin plus an optional aminoglycoside of choice, with the addition of intravenous (IV) ceftaroline fosamil, and will be given to all patients. Ceftaroline fosamil will be given at a dose of 6 mg/kg IV over 60 ( $\pm$  10) minutes every 8 hours (q8h) ( $\pm$  1 hour). If the presence of an organism that requires treatment with ampicillin cannot be excluded, then the use of IV ampicillin for the first 48 hours is mandatory. If the result of additional microbiology, polymerase chain reaction or other investigations, indicate that ampicillin during the first 48 hours of treatment is not required, then its use is at the discretion of the investigator.

The study design is described in the Study Diagram (Figure 1). Patient participation will require up to 49 days (up to 14 days of treatment plus up to 35 days of safety follow-up). The total duration of study therapy is 48 hours (minimum) to 14 days (maximum). Hospitalization is required during IV study therapy. Baseline assessments for study eligibility will occur within 36 hours before the first dose of study therapy.

Procedures will be performed according to the Study Plan in Table 1. Safety assessments will be done throughout the study. Between Day 2 and Day 14, 2 blood samples will be collected for PK analysis. The efficacy of ceftaroline fosamil will be evaluated based on the clinical outcome (clinical cure, clinical failure or indeterminate) at end of therapy (EOT; within 24 hours after completion of last infusion) and test-of-cure (TOC; 8 to 15 days after the last dose of study therapy) assessments. The Safety Follow-up (SFU) assessments will occur 28 to 35 days after the last dose of study therapy. Adverse events (AEs) will be followed up in the study until SFU.

A patient who is prematurely discontinued from study therapy administration for any reason will have EOT assessments conducted and undergo subsequent safety assessments at TOC and SFU per protocol.

- If a patient is prematurely discontinued from study therapy due to an adverse event and the clinical signs and symptoms of sepsis have resolved completely or improved such that no further antibacterial therapy is necessary, the patient will be assessed as a clinical cure at EOT and reassessed at TOC.
- If a patient is prematurely discontinued from study therapy due to a study therapyrelated AE and requires alternative non-study antibacterial for treatment for LOS, the patient will be assessed as a clinical failure (or indeterminate, if the patient discontinued before minimum treatment duration) at EOT and TOC.
- If a patient is prematurely discontinued from study therapy administration (at any time after the required minimum treatment duration of 48 hours) due to insufficient therapeutic effect, the patient will be assessed as a clinical failure on the day of discontinuation (ie, EOT) and at all subsequent evaluation time points.

A patient who is withdrawn completely from this study will undergo, if possible, EOT assessments per protocol on the day of withdrawal. Patients withdrawn from the study will not undergo subsequent TOC efficacy assessments. Patients who are withdrawn from the study and have not been assessed as clinical failure will be assessed as indeterminate for all remaining scheduled clinical assessments. Patients withdrawn from therapy and assessed as a clinical cure at EOT will undergo subsequent TOC efficacy assessments, if possible.

An external Data Safety Monitoring Board (DSMB) will review data on a regular basis to assess the safety of all patients enrolled in this and other ongoing pediatric studies of

ceftaoline fosamil. The scope of the DSMB and the data to be provided to them is documented in a separate DSMB charter.

Figure 1 Study Diagram



Abbreviations: EOT-end of therapy. ICF-informed consent. IV-intravenous. PK-pharmacokinetic. SFU-safety follow-up. TOC-test of cure.

An external Data and Safety Monitoring Board (DSMB) will be established to reviews a fety data from this study and other ongoing pediatric studies of ceftaroline fosamil on a regular basis to ensure safety of all subjects enrolled

\* IV ampicillin and optional aminoglycoside will be given as per standard of care. If the presence of an organism that requires treatment with ampicillin cannot be excluded, then the use of IV ampicillin for the first 48 hours is mandatory. If the result of additional microbiology, polymerase chain reaction or other investigations, indicate that ampicillin during the first 48 hours of treatment is not required, then its use is at the discretion of the investigator

\*\* Patients will be randomly assigned to PK schedule using IXRS

Table 1 Study Plan

| | | | | Tr | eat | ment pe | eriod | Follow-up | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment or Procedure | | D !! | Study Days* | | | | | | |
| | | Baseline | 1 | | | 4-14 | EOT b | TOC° | SFU <sup>d</sup> |
| | Written informed consent | X | | | | | | | |
| | Inclusion/exclusion criteria <sup>e</sup> | X | | | | | | | |
| | Medical history (including antepartum/peripartum period) | X | | | | | | | |
| | Adverse event review (AEs and SAEs) | X | X | X | X | X | X | X | X |
| | Prior and concomitant medications <sup>f</sup> | X | X | X | X | X | X | X | X |
| | Length | X | | | | | | | |
| ical | Weight | X | X | X | X | X | X | X | X |
| Clinical | Physical examination | X | X | X | X | X | X | X | |
| | Vital signs and oxygen saturation <sup>g</sup> | X | X | X | X | X | X | X | X |
| | Clinical outcome | | | | | | X | X | |
| | Record adjunctive therapeutic procedures (if performed) | | X | X | X | X | X | X | |
| | CXR, CT scan, or other imaging tests <sup>h</sup> | | | | | X <sup>j</sup> | ' | • | |
| | CBC with differential <sup>i</sup> | X | | | X | | X | X <sup>j</sup> | X <sup>j</sup> |
| | Chemistry panel <sup>i</sup> | X | | | X | | X | X <sup>j</sup> | X <sup>j</sup> |
| ory | Base excess | | • | Х | Z <sup>j</sup> | | | | |
| Laboratory | CRP and Procalcitonin <sup>i</sup> | | $X^{j}$ | | | | | | |
| Lab | Urinalysis | X | | | X | | X | X <sup>j</sup> | |
| | Urine output | X <sup>k</sup> | X | X | X | | X <sup>j</sup> | | |
| | CSF | | Xi | | | | | | |
| | Assignment to PK schedule <sup>1</sup> | X | | | | | | | |
| PK | PK blood sample <sup>m</sup> | | | | | X | | | |
| Ъ | CSF sample (if collected per standard of | | | | | | | | |
| care) & matching blood sample <sup>n</sup> | | X | | | | | | | |
| | Blood culture | | $X^{j}$ | | | | | | |
| Micro | Urine culture | | X <sup>j</sup><br>X <sup>j</sup> | | | | | | |
| Ψį | CSF culture | | | | | | | | |
| | Other specimen or tissue cultures | | | | | X <sup>j</sup> | | | |
| | Administration of study therapy | | X | X | X | X | X | | |

Abbreviations: AEs=adverse events; CBC=complete blood count; CRP=C-reactive protein; CSF=cerebrospinal fluid; CT=computed tomography; CXR=chest radiograph; EOT=End-of-Therapy; MRI=magnetic resonance imaging; PK=pharmacokinetic; SAEs=serious adverse events; SFU=Safety Follow-up; TOC=Test-of-Cure.

- a. Conduct Baseline assessments within 36 hours before first dose of study therapy.
- b. Conduct EOT assessments within 24 hours after the last dose of study therapy. Study therapy may or may not be given on the same calendar day as EOT assessments; administration should be as for days 4-14.
- c. Conduct TOC assessments 8 to 15 days after the last dose of study therapy.
- d. Conduct SFU assessments, preferably in person, 28 to 35 days after the last dose of study therapy. The SFU may be conducted via telephone for any patient who has not experienced clinical relapse, did not have ongoing AEs or SAEs at TOC, or did not develop AEs or SAEs since TOC. If symptoms of relapse or new AEs or SAEs are noted, or at the discretion of the investigator, the patient should be immediately scheduled for an in-person visit. If the visit is in-person, weight, vital signs and oxygen saturation should be recorded. If a patient was previously assessed as a clinical failure, only safety assessments will be performed.
- e. Refer to the inclusion criteria (Section 3.1 of the study protocol) for the recommended definitions of clinical and laboratory inclusion criteria.
- f. For patients who are being breast fed, record all medications taken by the lactating mother for 3 days before first dose of study therapy through SFU.
- g. Postbaseline, record highest and lowest postdose temperature measurements.
- h. At baseline, record results of CXR, CT scan, or other imaging tests (eg, echocardiogram, CT, MRI, sonography) if performed within 72 hours before first dose of study therapy.
- i. Refer to the inclusion criteria (Section 3.1 of the study protocol) for list of tests. Recommended to repeat at least every 7 days. If immature neutrophils are available, calculate I/T neutrophil ratio using the formula: I/T ratio=Immature cells/Total (mature+immature).
- j. If clinically indicated.
- k. For patients who have been hospitalized for ≥8 hours, calculate urine output over the last 8 hour period.
- 1. Patients will be randomly assigned (1:1) to one of the following PK sample collection schedules collected after any dose between the end of the 4th infusion of ceftaroline fosamil and before EOT or Study Day 14 (whichever is earlier):
  - PK Schedule 1: at the end of the ceftaroline fosamil infusion (± 5 minutes) and 3 to 4 hours after the end of the infusion
  - PK Schedule 2: 15 minutes to 2 hours after the end of the ceftaroline fosamil infusion and 5 to 7 hours after the end of the infusion (before the start of the next infusion).
- m. PK blood samples are NOT to be drawn if the patient received a blood or blood component transfusion within the past 24 hours. For patients who are at risk from additional blood loss, collection of PK samples will require assessment by the investigator.
- n. Matching blood sample to be collected only if 2 PK blood samples have not been collected already. The matching blood sample replaces one of the PK samples, so that the total number of PK samples does not exceed 2.

# 1.3 Number of patients

The primary objective of this study is to evaluate safety and tolerability of ceftaroline fosamil in neonates and young infants aged 7 to <60 days with LOS and the study is not powered for inferential statistical analysis. The sample size (24 patients; 3 cohorts of 8 patients) is considered adequate to evaluate the safety of ceftaroline fosamil in neonates and young infants with LOS.

#### 2. ANALYSIS SETS

# 2.1 Definition of analysis sets

Figure 2 shows the relationship among different analysis sets graphically. The analysis of data will be based on different analysis sets according to the purpose of analysis, ie, for safety, efficacy, etc.

Intent-to-Treat (ITT) All subjects Microbiological ITT (Micro-ITT) Subjects who have one or more potentially Safety causative baseline pathogens identified Received any amount of ceceftaroline fosamil Pharmacokinetic (PK) Received a known amount of ceftaroline fosamil and has ≥1 PK sample Modified Intent-to-Treat (MITT) Meets minimal disease criteria of LOS (excluding subjects with confirmed in fection with a resistant pathogen known to be resistant to ceftaroline fosamil; or confirmed fungal, parasitic, or viral pathogen as the sole cause of infection).

Figure 2 Study Analysis Sets

### 2.1.1 Intent-to-treat Analysis Set

The Intent-to-treat (ITT) Analysis Set will consist of all enrolled patients for whom informed consent form (ICF) was signed.

#### 2.1.2 Safety Analysis Set

The Safety Analysis Set will be a subset of the ITT Analysis Set and will include all patients who received any amount of ceftaroline fosamil.

#### 2.1.3 Modified Intent-to-Treat Analysis Set

The Modified Intent-to-treat (MITT) Analysis Set will include all patients who received any amount of ceftaroline fosamil and who met minimal disease criteria of LOS as described in the protocol inclusion criteria (diagnosis of sepsis within 36 hours before enrolment, defined as the presence of at least 2 clinical criteria and at least 1 laboratory criteria in the presence of or as a result of suspected or proven bacterial infection that requires IV antibiotic therapy). Patients with confirmed infection at baseline with a pathogen known to be resistant by CLSI methodologies and interpretive criteria (M100-S-28) to the study therapy received will be excluded. Patients with a confirmed fungal, parasitic, or viral pathogen as the sole cause of infection will also be excluded (Appendix A).

#### 2.1.4 Microbiological Intent-to-Treat Analysis Set

The Microbiological Intent-to-treat (Micro-ITT) Analysis Set will include all ITT subjects who have one or more potentially causative baseline pathogens identified.

#### 2.1.5 Pharmacokinetic (PK) Analysis Set

The PK Analysis Set will include all patients who received a known amount of ceftaroline fosamil, were randomized to a PK sample collection schedule, and had at least 1 PK sample collected.

#### 2.2 Protocol deviations

Per PRA processes all important protocol deviations (PDs) as identified in the protocol deviation guidance document will be tracked and entered into the Clinical Trials Management System (CTMS). The study team will conduct ongoing reviews of PD data from CTMS throughout the study. Protocol deviations that the study team considers not to be important will not be tabulated or listed. Important protocol deviations will be verified as part of the final data review before database lock.

#### 3. PRIMARY AND SECONDARY VARIABLES

For the calculation or derivations of the variables in this section, baseline will be defined as the last non-missing value before the start of study therapy. Change from baseline variables will be calculated for clinical laboratory tests and vital signs parameters as the post-treatment value minus the value at baseline. The visit windows for EOT, TOC, and SFU are defined in Table 2 for efficacy analyses.

Study days are to be calculated starting from the onset of the first dose of study therapy, in 24-hour increments. If a date is prior to the first study therapy dose date (eg, date of LOS diagnosis, prior medication start date) then the study day will be calculated as (past date – first

study therapy dose date); if the assessment date is on or after the first study therapy dose date then the study day will be calculated as (assessment date – first study therapy dose date + 1). Durations in days will be calculated as (end date – start date +1).

Table 2 Visit Windows for EOT, TOC, and SFU

| Visit | Protocol-defined Window |
|---|---|
| End of IV therapy (EOT) | Within 24 hours of completion of the last infusion of study drug |
| Test of cure (TOC) | 8 to 15 days after the last dose of study drug |
| Safety follow-up (SFU) | 28 to 35 days after the last dose of study drug |

NB. Since there is no per protocol population defined for this study, scheduled visits will be used for MITT analyses and derived analysis windows will not be evaluated.

For analyses purposes, nominal visit data was used.

# 3.1 Primary outcome variables

### 3.1.1 Safety variables

The safety analysis will be performed using the Safety Analysis Set. Safety parameters include AEs, serious adverse events (SAEs), deaths, clinical laboratory parameters (eg, complete blood count [CBC] with differential, chemistry panel), and vital signs.

No imputation on missing data will be undertaken for safety parameters.

#### 3.1.1.1 Adverse events (AE) variables

An AE is the development of any new undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (eg, nausea, chest pain), signs (eg, tachycardia, enlarged liver), or the abnormal results of an investigation (eg, laboratory findings). In clinical studies, an AE can include an undesirable medical condition occurring at any time, even if no study therapy has been administered. All AEs will be classified using the Medical Dictionary for Regulatory Activities (MedDRA) version 12.0 or higher.

The term AE is used to include both serious and nonserious AEs. Each AE will be graded for intensity (mild, moderate, severe). If intensity is missing it will be presented as such in the corresponding Tables. Each AE will be assessed for relationship to the study therapy (yes, no) as well. If relationship to study therapy is missing it will be presented as such in the corresponding Tables.

Adverse events will be collected from the time the parent(s)/legal guardian/legally acceptable representative provides informed consent throughout the treatment period up to and including the SFU visit in the study. AEs occurring after the start of administration of the first dose of study therapy or AEs that started prior to treatment and worsened on treatment up to and including the SFU visit will be summarised.

Adverse events of special interest (AESI) will be selected by subsetting MedDRA preferred terms from Pseudomembranous colitis Standard MedDRA Query (SMQ narrow), Anaphylactic reaction (SMQ narrow), Angioedema (SMQ narrow), and Malignancies (SMQ

narrow). The MedDRA preferred terms identifying the AESI were provided by Pfizer, see Appendix C.

#### Serious adverse events variables

A SAE is an AE occurring during any study phase (ie, treatment, follow-up), that fulfils one or more of the following criteria:

- Results in death
- Is immediately life threatening
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity
- Is a congenital abnormality or birth defect
- Is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above
- Is any suspected transmission via a medicinal product of an infectious agent.

SAEs will be collected from baseline throughout the treatment period up to and including the SFU visit in the study. SAEs occurring in a subject after the active collection period has ended are reported to Pfizer Safety if the investigator becomes aware of them; at a minimum, all SAEs that the investigator believes have at least a reasonable possibility of being related to investigational product must be reported to Pfizer Safety. SAEs reported after the active collection period will be reported in the Pfizer Safety database only, not in the clinical database.

Analysis of SAEs will focus on treatment-emergent SAEs which will be those occurring after the start of administration of the first dose of study therapy or SAEs that started prior to treatment and worsened on treatment.

#### 3.1.1.2 Death

For any patients who die during the study, date and time of death, autopsy yes/no, and primary and secondary cause of death will be collected.

#### 3.1.1.3 Clinical laboratory variables

The safety laboratory parameters presented in Table 3 will be measured.

 Table 3
 Laboratory safety variables

| Chemistry panel | CBC and differential | Urinalysis |
|---|---|---|
| Albumin | Haematocrit | Bilirubin |
| Alkaline phosphatase | Haemoglobin | Blood |
| Alanine aminotransferase | Red Blood Cell count | Glucose |
| Aspartate aminotransferase | White Blood Cell count | Protein |
| Bilirubin, total and direct | Eosinophils <sup>c</sup> | рН |
| Blood urea nitrogen | Lymphocytes <sup>c</sup> | Specific Gravity |
| Urea | Monocytes <sup>c</sup> | Colour |
| Calcium | Neutrophils <sup>c</sup> | Appearance |
| Chloride | Platelets | Nitrite |
| Creatinine <sup>a</sup> | Immature granulocytes <sup>c</sup> | Urobilinogen |
| Glucose, nonfasting <sup>a</sup> | Metamyelocytes <sup>c</sup> | Leukocyte esterase |
| Potassium | Myelocytes <sup>c</sup> | |
| Sodium | Promyelocytes <sup>c</sup> | |
| Bicarbonate (HCO <sub>3</sub> ) <sup>b</sup> | Blasts <sup>c</sup> | |
| Lactate Dehydrogenase <sup>b</sup> | | |
| $pH^b$ | | |
| C-reactive protein <sup>b</sup> | | |
| Procalcitonin <sup>b</sup> | | |

<sup>&</sup>lt;sup>a</sup> Required for eligibility.

Hematology and chemistry will be performed at every visit or as clinically indicated. Urinalysis, 8-hour urine output if available, and CSF samples will be collected through the TOC visit. If available, base excess (BE) will be calculated from blood gases, and C-reactive protein (CRP) and procalcitonin will be assessed during the treatment period only.

Système International units will be reported for all analytes. Local laboratory upper limit of the normal range (ULN) and lower limit of the normal range (LLN) values for laboratory parameters will be applied for safety data in this study. No ULN or LLN are defined for vital signs parameters in the pediatric setting. Selected potentially clinically significant (PCS) laboratory results will be defined; see Appendix B for a list of PCS laboratory results.

#### 3.1.1.4 Vital signs variables

Vital signs variables include weight, heart rate, blood pressure (systolic and diastolic), respiratory rate, and temperature will be assessed at every scheduled clinical visit. Highest and lowest daily temperature will be monitored as well. In addition, length will be collected at baseline only.

For heart rate and blood pressure measurements at baseline, at least 2 measurements will be taken during a 30 minute period; the mean of all measurements will be utilized for analysis.

b Test not mandatory for eligibility if other eligibility criteria are met.

<sup>&</sup>lt;sup>c</sup> Absolute count and/or %.

### 3.1.1.5 Other safety variables

Other safety variables include:

- Physical exam by body system (general appearance, skin, head and neck, lymph nodes, musculoskeletal/extremities, cardiovascular, respiratory, abdomen, and neurological) through TOC, with specification of baseline and new/aggravated abnormalities
- Imaging study results (chest radiograph [CXR], computed tomography [CT] scan, or other radiology) through TOC including location, type of examination, result normal/abnormal, and description of abnormal findings
- Adjunctive therapeutic procedures related to infections variables through TOC including procedure, procedure type, other (specify), start date and time, stop date and time, and reason for procedure.

# 3.2 Secondary outcome variables

#### 3.2.1 Efficacy variables

#### 3.2.1.1 Clinical response variable at EOT and TOC

Efficacy outcome measures will include clinical response at EOT and TOC. The clinical outcome categories at EOT are defined in Table 4 below and the clinical outcome categories at TOC as defined in Table 5 below. A favourable outcome is clinical cure.

Table 4 Clinical outcome categories at End-of-Therapy

| Outcome | Definition |
|---|---|
| Clinical Cure | Resolution of all acute signs and symptoms of LOS or improvement to such an extent that no further antibacterial therapy is required |
| Clinical Failure | <ul> <li>Subjects who received ≥48 hours of study treatment and meet any of the following: <ul> <li>Discontinuation of study therapy due to insufficient therapeutic effect, including persistence, incomplete clinical resolution, worsening in signs and symptoms of LOS, or isolation of a resistant pathogen that requires alternative nonstudy antibacterial therapy</li> <li>Discontinuation of study therapy due to a study therapy-related AE and requirement for alternative nonstudy antibacterial therapy for LOS</li> <li>Death in which LOS is contributory</li> </ul> </li> </ul> |
| Indeterminate | <ul> <li>Study data are not available for evaluation of efficacy for any reason, including:</li> <li>Death in which LOS is clearly noncontributory</li> <li>Lost to follow-up</li> <li>Extenuating circumstances precluding classification as a cure or failure</li> <li>Diagnosis of CNS infection, osteomyelitis, endocarditis, or NEC at any time after enrolment</li> <li>Received &lt;48 hours of study therapy</li> </ul> |

Abbreviations: AE=adverse event; CNS=central nervous system; LOS=late-onset sepsis; NEC=necrotizing enterocolitis.

Table 5 Clinical outcome categories at Test-of-Cure

| Outcome | Definition |
|---|---|
| Clinical Cure | Resolution of all acute signs and symptoms of LOS or improvement to such an extent that no further antibacterial therapy is required |
| Clinical Failure | Subjects who received ≥48 hours of study treatment and meet either of the following criteria: • Incomplete resolution or worsening of LOS signs or symptoms or development of new signs or symptoms, or isolation of a resistant pathogen requiring alternative nonstudy antibacterial therapy • Death in which LOS is contributory |
| Indeterminate | <ul> <li>Study data are not available for evaluation of efficacy for any reason, including:</li> <li>Death in which LOS is clearly noncontributory</li> <li>Lost to follow-up</li> <li>Extenuating circumstances precluding classification as a cure or failure</li> <li>Diagnosis of CNS infection, osteomyelitis, endocarditis, or NEC at any time after enrolment</li> <li>Received &lt;48 hours of study therapy</li> </ul> |

Abbreviations: CNS=central nervous system; LOS=late-onset sepsis; NEC=necrotizing enterocolitis.

Per-patient clinical response at TOC will be derived from clinical outcome (ie, investigator assessment) of clinical cure, clinical failure, or indeterminate at EOT and TOC as shown in Table 6 below.

Missing values may occur due to failure to record a response at TOC due to earlier clinical failure. An outcome of clinical failure at EOT will be carried forward to TOC. Missing values may occur due to premature discontinuation from study therapy administration. Patients who were prematurely discontinued from study therapy administration for any reason will have EOT assessments conducted (see Section 1.2) and will have per-patient clinical response at TOC derived according to the rules in Table 6. Unrelated deaths will be assessed as indeterminate for all remaining scheduled clinical assessments. Deaths occurring after TOC will not retrospectively change the TOC outcome (ie, if a patient was a clinical cure at TOC but died after TOC their clinical response at TOC remains clinical cure).

Table 6 Derivation of clinical response at TOC

| <b>EOT Outcome</b> | TOC Outcome | Clinical Response at TOC |
|--------------------|------------------|--------------------------|
| Clinical Cure | Clinical Cure | Clinical Cure |
| | Clinical Failure | Clinical Failure |
| | Indeterminate | Indeterminate |
| | Missing | Indeterminate |
| Clinical Failure | Clinical Cure | Clinical Failure |
| | Clinical Failure | Clinical Failure |
| | Indeterminate | Clinical Failure |
| | Missing | Clinical Failure |
| Indeterminate | Clinical Cure | Clinical Cure |
| | Clinical Failure | Clinical Failure |
| | Indeterminate | Indeterminate |
| | Missing | Indeterminate |

The proportion of MITT Analysis Set patients with a clinical cure will be defined using the following formula:

Number of patients with clinical response at TOC=clinical cure

(Number of patients with clinical cure + Number of patients with clinical failure + Number of patients with indeterminate)

The proportion of MITT Analysis Set patients with clinical failure and with indeterminate clinical response will be calculated analogously. For proportion of patients with clinical cure, clinical failure, and indeterminate, indeterminate or missing assessments will be included in the denominator for calculation of the proportions for the MITT Analysis Set.

# 3.2.1.2 Per-pathogen and per-patient microbiological response variables at EOT and TOC

The per-pathogen microbiological outcome categories for pathogens identified at baseline are defined in Table 7. Local microbiology data will only be used when central data is not available, for example, samples were not sent to the central laboratory for processing. Please see section 3.3.1.3 for further details.

Table 7 Per-pathogen microbiological response categories

| Microbiological | Definition | Response |
|---|---|---|
| Response <sup>a</sup> | | Category |
| Eradication | Source specimen demonstrated absence of the original baseline pathogen | Favorable |
| Presumed eradication | Source specimen was not available to culture and the patient was assessed as a clinical cure | Favorable |
| Persistence | Source specimen demonstrates continued presence of the original baseline pathogen | Unfavorable |
| Presumed persistence | Source specimen was not available to culture and the patient was assessed as a clinical failure | Unfavorable |
| Indeterminate | Source specimen was not available to culture and<br>the patient's clinical outcome was assessed as<br>indeterminate | Indeterminate |

<sup>&</sup>lt;sup>a</sup> For patients who were clinical failures before TOC, the microbiological outcome will be carried forward to TOC and will be determined based on the cultures and/or clinical outcome at the time of the early clinical failure determination.

Similarly, per-patient microbiological response will be categorized as favorable, unfavorable, or indeterminate as follows. Per-patient microbiological response at EOT and TOC will be derived programmatically based on individual outcomes for each baseline pathogen. In order for a patient to have a favorable per-patient microbiological response, the outcome for each baseline pathogen must be favorable (eradicated or presumed eradicated) at that time point. This includes results of blood cultures, urine cultures, CSF cultures or other specimen cultures at the time point. If the outcome for any baseline pathogen from any culture is unfavorable (persistence or presumed persistence) at that time point, the patient will be considered to have an unfavorable per-patient microbiological response. If there is an indeterminate per-pathogen microbiological response at the time point (ie, no culture result available and patient's clinical outcome was indeterminate), the patient will be considered to have an indeterminate per-patient microbiological response. For per-patient microbiological response at TOC visit, the above definition is only applicable to patients who are not clinical failures at EOT. Patients who are clinical failures at EOT will have the corresponding per-patient microbiological outcome determined from EOT cultures and carried forward to TOC. If no EOT culture is available for patients who are clinical failures at EOT, then the microbiological outcome at TOC will be presumed persistence. Otherwise, the microbiological outcome at TOC will be determined from cultures obtained within the TOC visit window. If no culture is available in the TOC window, then the microbiological outcome at TOC will be presumed from the clinical response at TOC (if clinical cure, the microbiological outcome will be presumed eradication; if clinical failure, the microbiological outcome will be presumed persistence; if clinically indeterminate, the microbiological outcome will be indeterminate).

#### 3.2.2 Pharmacokinetic variables

Two PK samples will be obtained at steady state from at least 20 patients to determine the population pharmacokinetics of ceftaroline fosamil, ceftaroline, and ceftaroline M-1 in this patient population. If CSF sample collection is expected per standard of care, PK blood samples should be collected at the time of CSF collection as a matching sample (see section

5.4.1 of the protocol). The total number of PK blood samples will not exceed 2. After the 2 PK blood samples have been collected, any portion of a CSF sample (collected as part of standard of care) not required for the patient's medical care should be retained for PK analysis.

Pharmacokinetic variables include actual sample collection times and plasma concentrations of ceftaroline fosamil, ceftaroline, and ceftaroline M-1 at each time point. If available, concentrations of ceftaroline and ceftaroline M-1 in cerebrospinal fluid (CSF) will be reported.

Plasma concentrations of ceftaroline fosamil, ceftaroline and ceftaroline M-1 will be listed by age cohort.

Covance Laboratories, using appropriate bioanalytical methods will determine plasma concentrations of ceftaroline fosamil, ceftaroline, and ceftaroline M-1.

#### 3.3.1 Demographic and baseline characteristic variables

#### 3.3.1.1 Demographic variables

Demographic variables include age (days), sex, race, and ethnicity. Age (days) will be calculated as (date of informed consent - date of birth + 1).

# 3.3.1.2 Surgical and medical history variables including antepartum/ peripartum period

Surgical history variables include procedures, study day of procedure start date, and current medication yes/no. Medical history variables include diagnosis, study day of condition start date and duration of condition (see Section 3 for calculation of study day and duration), status (past or current), and any current medication yes/no. Surgical and medical histories will be coded using MedDRA Version 12.0 or higher.

# 3.3.1.3 Baseline microbiological assessment variables for blood, CSF, urine, and other specimens

Identification of pathogens and susceptibility results will be recorded by both the local microbiology laboratory and the central reference laboratory. The identification and susceptibility results of the central microbiology reference laboratory will be regarded as definitive, if after re-testing, any discrepancies noted are not resolved. In the circumstance that the central lab could not isolate any organism from the submitted specimen, the local lab result will be used for organism identification (not including a result of "No Growth" at the central laboratory, which should be reported).

Microbiological assessments at baseline include collection data, culture data, antibiotic susceptibility data, and gram stain data:

 Collection data: specimen collected yes/no, type of specimen, reason for no specimen, specify if attempt made but unable to obtain, collection date and time and specimen acquisition method

- Culture data: specimen work up performed by, culture outcome, culture source location, laboratory name and identifier, pathogen type, isolate identification, isolate classification, isolate quantitation for 1 μL, 5 μL, 10 μL plates (for urine specimens only), isolate sent to central lab yes/no, reason if no specimen sent to central laboratory, accession identifier primary and secondary
- Antibiotic susceptibility data: local susceptibility tested yes/no, isolate identification, antibiotics tested, susceptibility, susceptibility criteria and susceptibility method
- Gram stain data: gram stain done yes/no, specify if no gram stain done and gram stain results, for example, epithelial cell results, etc.

## 3.3.2 Definition of prior and concomitant medication

Any medications (non-antimicrobial, antimicrobial, parenteral nutrition and blood/blood-component transfusions) taken by the patient between 7 days prior to study entry (or taken by the lactating mother of breast fed patients within 3 days prior to study entry) and prior to the first dose date of study therapy received will be considered prior medication. Any medication taken by the patient (or by the lactating mother of breast fed patients) at any time between dates of the first dose (including the date of the first dose) of study therapy through the TOC visit, inclusive, will be considered concomitant medication. Any medication started prior to the study entry and ended/ongoing up to the TOC will be considered as both prior and concomitant medication.

If any medications reported are not able to be determined as prior medications or concomitant medications due to missing or partial start dates and/or stop dates, the following imputation rules will be implemented:

- If the year is present but the month and day are missing, then 01JAN will be imputed for the start date and 31DEC for the stop date.
- If the year and month are present but the day is missing, then 01 will be imputed for the start date and the last day of the month for the stop date.

If both stop/start years are missing or both stop/start dates otherwise cannot be imputed, then the date will be treated as missing and the medication will be treated as both prior and concomitant medications.

#### 3.3.3 Exposure and Compliance variable

Exposure to the study therapy will be calculated as the difference between the last study therapy date and the first study therapy date converted to days plus 1 day. Any partial infusion will be considered as a complete infusion for the purpose of exposure, and the relevant details will be listed.

Compliance will be calculated as the sum of the actual infusions over all doses/expected infusions over all doses)\*100.

#### 4. ANALYSIS METHODS

# 4.1 General principles

All analyses will use SAS<sup>®</sup> version 9.1.3 or higher. Summary tables will be organized by age cohort and overall. All available data for each analysis set will be used in the analyses, and a subset of key safety, efficacy, and PK data will be included in listings. No statistical hypothesis testing will be performed. Confidence intervals (CI) will be two-sided 95% CIs.

Unless otherwise noted, categorical data will be presented using counts and percentages with the denominator for percentages being the number of patients in the analysis set by age cohort. Percentages will be rounded to one decimal place; except 0% and 100% will be displayed without any decimal places and percentages will not be displayed for zero counts. Continuous variables will be summarized using the number of observations (n), mean, SD, median, minimum, and maximum. The minimum and maximum values will be displayed to the same level of precision as the raw data, the mean and median to a further decimal place and the SD to two additional decimal places.

Imputation of missing data will be performed as described within this document (see Section 3.2.1 for imputation of efficacy data at EOT and TOC and Section 3.3.2 for imputation of partial dates for prior and concomitant medication). Visit windowing will be performed as described in Section 3.

Baseline summaries will utilize the ITT and MITT Analysis Sets. Study therapy exposure, concomitant medication, and safety analyses will utilize the Safety Analysis Set. Efficacy analyses of clinical outcome and microbiological response will utilize the MITT and Micro-ITT Analysis Sets. PK analyses will utilize the PK Analysis Set. All data will be listed.

#### 4.1.1 Data quality

The clinical database will be cleaned prior to analysis; see PRA Clinical Informatics Plan for details. Beyond the data screening built into the PRA Clinical Informatics Plan, the PRA programming of analysis datasets, tables, figures, and listings (TFLs) will provide additional data screening.

Review of a pre-freeze TFL run on clean patients and a post-freeze TFL run on the frozen database will allow for further data screening prior to lock. The post-freeze TFL will be discussed with Pfizer in a data review meeting to identify any final data issues and seek corrections prior to database lock. The PRA statistician and Pfizer must approve database lock.

PRA's goal is to ensure that each TFL delivery is submitted to the highest level of quality. Our quality control procedures will be documented separately in the study-specific clinical programming quality control plan.

# 4.2 Analysis methods

#### 4.2.1 Patient disposition

The number and percentage of patients enrolled and treated with study therapy, along with the number and percentage of treatment completers, premature discontinuations from study

therapy administration, and withdrawals from the study will be provided overall and within each age cohort based for all patients, ie, all subjects who signed informed consent.

Disposition details for subjects who discontinued from the study and from study therapy; and those who completed the study will be listed for all patients.

The number of patients in each analysis set and the reasons for exclusion from analysis sets will be listed and summarized for the ITT Analysis Set.

#### 4.2.2 Protocol deviations

A table of important PDs will be presented overall and by age cohort for the ITT Analysis Set. See Section 2.2 for details, including determination of importance.

Important PDs will be displayed in a data listing by age cohort and patient.

#### 4.2.3 Demographics and baseline characteristics

Demographics data defined in Section 3.3.1 will be summarized for the ITT, MITT and Micro-ITT Analysis Set by age cohort and overall. Baseline length (cm) and weight (kg) will be tabulated.

Relevant surgical and medical history (past and current) including antepartum/peripartum period will be summarized by MedDRA System Organ Class and preferred term, both by age cohort and overall for the ITT Analysis Set.

The number and percentage of patients with baseline pathogens (Genus and species) by specimen type (blood, CSF, urine, and other specimens) will be summarized by age cohort and overall for the ITT, MITT and Micro-ITT Analysis Set.

Demographics and baseline characteristics, and relevant medical and surgical history data will be listed by age cohort and patient. Baseline culture data including susceptibility (susceptible, intermediate, resistant) and gram stain testing results will be listed by age cohort and patient for the ITT Analysis Set.

#### 4.2.4 Prior and concomitant medications

See Section 3.3.3 for definitions of prior and concomitant medications.

Medications received concomitantly with study therapy, categorized by anatomical therapeutic chemical classification and generic name according to the World Health Organization Drug Dictionary Enhanced (WHODDE, Version 20.0), will be summarized. The number and percentage of patients using at least one medication within each ATC Group and Generic Term will be displayed by age cohort and overall for the Safety Analysis Set. Prior medications will be summarized in an identical fashion. For lactating mothers, maternal prior and concomitant medications will be included in these summaries.

The duration of prior medications defined as the end date – start date +1, will also be summarized for each ATC Group and Generic Term and displayed by age cohort and overall for the ITT Analysis Set. In the event that prior medications had partial dates no imputation will be undertaken and consequently the duration of prior medication will be missing for any such records.

Prior and concomitant medication data will be listed for the ITT Analysis Set by age cohort and patient.

#### 4.2.5 Study therapy exposure and compliance

Duration of study therapy exposure in days for ceftaroline fosamil, optional ampicillin and optional aminoglycoside will be tabulated by age cohort and overall for the Safety Analysis Set and MITT population. In addition to standard summary statistics, quartiles for each patient and total treatment days for all patients will be shown.

Following protocol amendment 2 the dose of ceftaroline fosamil was changed from 4mg/kg to 6mg/kg. No summaries will be provided by the different ceftaroline fosamil doses, under the different versions of the protocol to which patients were enrolled.

Treatment compliance will be summarized as continuous data and categorically (<80%, 80-120%, >120% compliance) by age cohort and overall for the Safety Analysis Set and MITT population.

Ceftaroline fosamil exposure data, compliance data and administration details will be listed by age cohort and patient for the Safety Analysis Set.

#### 4.2.6 Safety analysis

### 4.2.6.1 Analysis of adverse events, serious adverse events, and deaths

The number and percentage of patients with AEs occurring after the start of administration of the first dose of study therapy, or AEs that started prior to treatment and worsened on treatment, up to the SFU visit will be summarized, i.e. treatment emergent(TE) AEs. The following summaries will be presented for the Safety Analysis Set:

- Overall summary of TEAEs by category (overall and by age cohort)
- Incidence of TEAEs by system organ class (SOC) and preferred term
- Incidence of TEAEs by SOC, preferred term, and maximum intensity
- Incidence of TEAEs by SOC, preferred term, and relationship to ceftaroline
- Incidence of TEAEs of special interest by SOC and preferred term
- Incidence of non-serious TEAEs by SOC and preferred term
- Incidence of TEAEs with fatal outcome by SOC and preferred term
- Incidence of all deaths
- Incidence of Serious TEAEs by SOC and preferred term
- Incidence of TEAEs leading to discontinuation of investigational product by SOC and preferred term

All AEs occurring prior to the first intake of ceftaroline will be listed for the Safety Analysis Set.

#### 4.2.6.2 Clinical laboratory safety assessment

Clinical laboratory data include hematology, chemistry, CRP, CSF, blood gas and base excess, urinalysis, and urine output. Descriptive statistics (including n, mean, SD, minimum, median, and maximum) of observed results and change from baseline will be presented for continuous clinical laboratory results by age cohort and overall for the Safety Analysis Set.

In addition, the following summaries at each applicable visit will also be provided by age cohort and overall:

- Shift tables showing the number of patients with changes from low, normal, or high values from baseline
- Shift tables showing the number of patients with urinalysis changes from baseline to each category (negative, trace, positive)
- The number and percentage of patients with abnormal values using the PCS criteria in Appendix B

Listings of values for each patient will be presented by age cohort with abnormal or out-ofrange values flagged. All laboratory results for each patient will be listed for the Safety Analysis Set.

#### 4.2.6.3 Weight, vital signs, and oxygen saturation results

Weight, vital signs (heart rate, blood pressure, respiratory rate, temperature) and oxygen saturation (measured by oximeter) will be summarized. Descriptive statistics (including n, mean, SD, minimum, median, and maximum) of observed results and change from baseline will be presented for continuous results by age cohort and overall for the Safety Analysis Set.

Listings of values for each patient will be presented by age cohort for the Safety Analysis Set.

#### 4.2.6.4 Other safety results

Data for physical examination by body system, imaging study results, and adjunctive therapeutic procedures related to infections will be included in ADaM datasets and presented in listings for the Safety Analysis Set.

#### 4.2.7 Efficacy analysis

#### 4.2.7.1 Clinical response

The number and percentage of patients with a clinical cure, clinical failure, and indeterminate clinical response at EOT and TOC will be tabulated overall and by baseline pathogen, overall and within each age cohort for the ITT, MITT and Micro-ITT Analysis Sets. A two-sided 95% CI for the observed clinical cure rate overall, within each cohort and overall will be constructed using the Jeffreys method. Sensitivity analyses will be conducted on the overall response excluding indeterminate responses.

Clinical outcome and derived response data will be listed by age cohort and patient for the ITT Analysis Set.

#### 4.2.7.2 Microbiological response

The number and percentage of patients with a favourable, unfavourable and indeterminate microbiological response at EOT and TOC will be tabulated overall, and by baseline pathogen (overall and within each age cohort) for the MITT and Micro-ITT Analysis Sets. A two-sided 95% CI for the observed microbiological favourable rate overall within each cohort and overall will be constructed using the Jeffreys method.

The number and percentage of pathogens with a favorable microbiological response (eradication, presumed eradication) at TOC will be tabulated by baseline pathogen and baseline ceftaroline MIC (overall and within each age cohort) for the MITT and Micro-ITT Analysis Sets.

All other microbiological data including microbiological responses by pathogen and by patient, susceptibility testing and gram staining will be listed by age cohort and patient for the ITT Analysis Set.

#### 4.2.8 Pharmacokinetics analysis

Ceftaroline plasma concentration data, along with other information including demographic data, will be combined with appropriate data from other clinical studies and analyzed using a population PK approach and reported separately.

PK schedule assignment data, sample collection data and plasma concentration data will be listed by age cohort and patient for the PK Analysis Set.

#### 5. APPENDICES

APPENDIX A Non-eligible pathogens

APPENDIX B Criteria for potentially clinically significant laboratory results

APPENDIX C Adverse Events of Special Interest

# Appendix A Non-eligible pathogens

 Table 2
 Pathogen Classifications for Study

| 1 able 2 Patnogen Classifications for Study | | |
|---|---|---|
| Always | Never | Sometimes |
| Enterobacteriaceae | ESBL phenotype positive | Enterococcus spp.* |
| | Enterobacteriaceae | |
| Staphylococcus aureus | | |
| | Other Enterobacteriaceae not | |
| Streptococcus spp. | susceptible to study drug received | |
| Coagulase-negative | Other non-Enterobacteriaceae | |
| staphylococci | Gram negative bacteria | |
| Streptococcus spp. | Non-fermentative Gram-negative | |
| (except viridans Streptococci) | bacteria including Pseudomonas | |
| ( P | spp. | |
| | SPP. | |
| | viridans Streptococci | |
| | ······································· | |
| | Anaerobes | |
| | Fungal pathogens (including yeast) | |
| | Parasitic pathogens | |
| | Viral pathogens | |
| | 1 0 | |

Table 1 represents the latest known list for pathogens susceptible to ceftaroline. If more data become available during the course of this study, then this list will be updated appropriately.

<sup>\*</sup> Based on investigator determination.

# Appendix B Criteria for Potentially Clinically Significant Laboratory Tests

| Category | Category<br>Parameter | Lower<br>Limit | Upper<br>Limit | Percent<br>decrease from | Percent increase from |
|---|---|---|---|---|---|
| TT , 1 | TT | .0.6. 1131 | . 10 11131 | baseline | baseline |
| Haematology | Haematocrit | < 0.6 x LLN | > 1.3 x ULN | > 25% | > 30% |
| | Haemoglobin | < 0.6 x LLN | > 1.3 x ULN | > 25% | > 30% |
| | Red Blood Cell | < 0.8 x LLN | > 1.3 x ULN | > 20% | > 30% |
| | count | 0.7.777 | | 500/ | 1000/ |
| | White Blood Cell | < 0.5 x LLN | > 2.0 x ULN | > 60% | > 100% |
| | count | | | | |
| | Eosinophils | N/A | > 4.0 x ULN | N/A | > 400% |
| | Lymphocytes | < 0.2 x LLN | > 2.2 x ULN | > 70% | > 100% |
| | (absolute count) | | | | |
| | Neutrophils | < 0.5 x LLN | > 2.2 x ULN | > 70% | > 100% |
| | (absolute count) | | | | |
| | Platelets | < 0.4 x LLN | > 2.0 x ULN | > 40% | > 100% |
| Haematology/ | International | < 0.5 x LLN | > 2.0 x ULN | > 50% | > 100% |
| Coagulation | normalized ratio | | | | |
| | Partial | < 0.5 x LLN | > 2.0 x ULN | > 50% | > 100% |
| | thromboplastin time | | | | |
| | Prothrombin Time | < 0.5 x LLN | > 2.0 x ULN | > 50% | > 100% |
| Chemistry | Albumin | < 0.6 x LLN | N/A | > 60% | N/A |
| | Alkaline | < 0.5 x LLN | > 3.0 x ULN | > 80% | > 300% |
| | phosphatase | | | | |
| | Alanine | N/A | > 3.0 x ULN | N/A | > 300% |
| | aminotransferase | | | | |
| | Aspartate | N/A | > 3.0 x ULN | N/A | > 300% |
| | aminotransferase | | | | |
| | Bilirubin, direct | N/A | > 2.5 x ULN | N/A | > 150% |
| | Bilirubin, total | N/A | > 2.5 x ULN | N/A | > 300% |
| | Bilirubin, indirect | N/A | > 2.5 x ULN | N/A | > 150% |
| | Blood urea | N/A | > 3 x ULN | N/A | > 300% |
| | nitrogen* | | | | |
| | Calcium | < 0.7 x LLN | > 1.3 x ULN | > 30% | > 30% |
| | Chloride | < 0.8 x LLN | > 1.2 x ULN | > 20% | > 20% |
| | Creatinine | N/A | > 2.0 x ULN | N/A | > 100% |
| | Glucose, nonfasting | < 0.6 x LLN | > 4.0 x ULN | > 40% | > 200% |
| | Potassium | < 0.8 x LLN | > 1.2 x ULN | > 15% | > 20% |
| | Sodium | < 0.85 x | > 1.1 x ULN | > 10% | > 10% |
| | | LLN | | | |
| | Lactate | < 0.4 x LLN | > 4.0 x ULN | > 60% | > 300% |
| | Dehydrogenase | , | | | |

PCS are based on P903-21 Study and consistent with Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November 2014 with grade 2 or greater laboratory abnormalities being considered PCS and Harriet Lane Handbook Version 19.

<sup>\*</sup> For sites that collect Urea instead of BUN, Urea will be converted to BUN using the following formula: Urea [mg/dL]/2.14 = BUN [mg/dL].

# **Appendix C Adverse Events of Special Interest**

| SMQ PTs taken from Anaphylactic reaction (SMQ) narrow | | |
|---|---|---|
| MedDRA v20.1 Preferred Term (PT) | | |
| Anaphylactic reaction Anaphylactic shock Anaphylactic transfusion reaction Anaphylactoid reaction | Anaphylactoid shock Circulatory collapse Dialysis membrane reaction Kounis syndrome | Shock Shock symptom Type I hypersensitivity |

| SMQ PTs taken from Angioedema (SMQ) narrow | | |
|---|---|---|
| MedDRA v20.1 Preferred Term (PT) | | |
| Allergic oedema | Idiopathic angioedema | Palatal oedema |
| Angioedema | Idiopathic urticaria | Palatal swelling |
| Circumoral oedema | Intestinal angioedema | Periorbital oedema |
| Conjunctival oedema | Laryngeal oedema | Pharyngeal oedema |
| Corneal oedema | Laryngotracheal oedema | Scleral oedema |
| Epiglottic oedema | Limbal swelling | Swelling face |
| Eye oedema | Lip oedema | Swollen tongue |
| Eye swelling | Lip swelling | Tongue oedema |
| Eyelid oedema | Mouth swelling | Tracheal oedema |
| Face oedema | Oculorespiratory syndrome | Urticaria |
| Gingival oedema | Oedema mouth | Urticaria cholinergic |
| Gingival swelling | Oropharyngeal oedema | Urticaria chronic |
| Gleich's syndrome | Oropharyngeal swelling | Urticaria papular |
| Hereditary angioedema | | F of the second |

| SMQ PTs taken from Malignancies (SMQ) narrow | | |
|---|---|---|
| MedDRA v20.1 Preferred Term (PT) | | |
| 5q minus syndrome | Gestational trophoblastic tumour | Ostectomy |
| Abdominal neoplasm | Gingival cancer | Osteosarcoma |
| Abdominal wall neoplasm | Glioblastoma | Osteosarcoma metastatic |
| Abdominal wall neoplasm malignant | Glioblastoma multiforme | Osteosarcoma recurrent |
| Acanthosis nigricans | Glioma | Otic cancer metastatic |
| Acinar cell carcinoma of pancreas | Gliomatosis cerebri | Ovarian cancer |
| Acinic cell carcinoma of salivary gland | Glioneuronal tumour | Ovarian cancer metastatic |
| Acquired thalassaemia | Gliosarcoma | Ovarian cancer recurrent |
| Acral lentiginous melanoma | Glossectomy | Ovarian cancer stage I |
| Acral lentiginous melanoma stage I | Glottis carcinoma | Ovarian cancer stage II |
| Acral lentiginous melanoma stage II | Glucagonoma | Ovarian cancer stage III |
| Acral lentiginous melanoma stage III | Good syndrome | Ovarian cancer stage IV |
| Acral lentiginous melanoma stage IV | Granular cell tumour | Ovarian clear cell carcinoma |
| Acrokeratosis paraneoplastica | Granulosa cell tumour of the testis | Ovarian dysgerminoma stage I |
| ACTH-producing pituitary tumour | Growth hormone-producing pituitary | Ovarian dysgerminoma stage II |
| Acute biphenotypic leukaemia | tumour | Ovarian dysgerminoma stage III |
## MedDRA v20.1 Preferred Term (PT)

Acute leukaemia Acute leukaemia in remission Acute lymphocytic leukaemia Acute lymphocytic leukaemia (in remission) Acute lymphocytic leukaemia recurrent Acute lymphocytic leukaemia refractory Acute megakaryocytic leukaemia Acute megakaryocytic leukaemia (in remission) Acute monocytic leukaemia Acute monocytic leukaemia (in remission) Acute myeloid leukaemia Acute myeloid leukaemia (in remission) Acute myeloid leukaemia recurrent Acute myelomonocytic leukaemia Acute promyelocytic leukaemia Acute promyelocytic leukaemia differentiation syndrome Acute undifferentiated leukaemia Adenocarcinoma Adenocarcinoma gastric Adenocarcinoma of appendix Adenocarcinoma of colon Adenocarcinoma of salivary gland Adenocarcinoma of the cervix Adenocarcinoma pancreas Adenoid cystic carcinoma Adenoid cystic carcinoma of external auditory canal Adenoid cystic carcinoma of salivary gland Adenosquamous carcinoma of the cervix Adenosquamous carcinoma of vagina Adenosquamous cell carcinoma Adenosquamous cell lung cancer Adenosquamous cell lung cancer recurrent Adenosquamous cell lung cancer stage 0 Adenosquamous cell lung cancer stage I Adenosquamous cell lung cancer stage Adenosquamous cell lung cancer stage Adenosquamous cell lung cancer stage IV Adrenal gland cancer Adrenal gland cancer metastatic Adrenal neoplasm Adrenocortical carcinoma Adult T-cell lymphoma/leukaemia Adult T-cell lymphoma/leukaemia recurrent Adult T-cell lymphoma/leukaemia

refractory

Haemangiopericytoma Haemangiopericytoma of meninges Haematological malignancy Haematopoietic neoplasm Haemorrhagic tumour necrosis Hairy cell leukaemia Hairy cell leukaemia recurrent Head and neck cancer Head and neck cancer metastatic Head and neck cancer stage I Head and neck cancer stage II Head and neck cancer stage III Head and neck cancer stage IV Hemicorporectomy Hemilaryngectomy Hemipelvectomy Hepatectomy Hepatic angiosarcoma Hepatic cancer Hepatic cancer metastatic Hepatic cancer recurrent Hepatic cancer stage I Hepatic cancer stage II Hepatic cancer stage III Hepatic cancer stage IV Hepatic neoplasm Hepatobiliary cancer Hepatobiliary cancer in situ Hepatobiliary neoplasm Hepatoblastoma Hepatoblastoma recurrent Hepatocellular carcinoma Hepatosplenic T-cell lymphoma HER-2 positive breast cancer HER-2 positive gastric cancer Hereditary leiomyomatosis renal cell carcinoma Hereditary papillary renal carcinoma Hidradenocarcinoma High frequency ablation High grade B-cell lymphoma Burkittlike lymphoma High grade B-cell lymphoma Burkittlike lymphoma recurrent High grade B-cell lymphoma Burkittlike lymphoma refractory High grade B-cell lymphoma Burkittlike lymphoma stage I High grade B-cell lymphoma Burkittlike lymphoma stage II High grade B-cell lymphoma Burkittlike lymphoma stage III High grade B-cell lymphoma Burkittlike lymphoma stage IV High intensity focused ultrasound High-grade B-cell lymphoma

Ovarian dysgerminoma stage IV Ovarian dysgerminoma stage unspecified Ovarian embryonal carcinoma Ovarian endometrioid carcinoma Ovarian epithelial cancer Ovarian epithelial cancer metastatic Ovarian epithelial cancer recurrent Ovarian epithelial cancer stage I Ovarian epithelial cancer stage II Ovarian epithelial cancer stage III Ovarian epithelial cancer stage IV Ovarian germ cell cancer Ovarian germ cell cancer stage I Ovarian germ cell cancer stage II Ovarian germ cell cancer stage III Ovarian germ cell cancer stage IV Ovarian germ cell choriocarcinoma Ovarian germ cell choriocarcinoma Ovarian germ cell choriocarcinoma stage II Ovarian germ cell choriocarcinoma stage III Ovarian germ cell choriocarcinoma stage IV Ovarian germ cell embryonal carcinoma stage I Ovarian germ cell embryonal carcinoma stage II Ovarian germ cell embryonal carcinoma stage III Ovarian germ cell embryonal carcinoma stage IV Ovarian germ cell endodermal sinus tumour Ovarian germ cell endodermal sinus tumour stage I Ovarian germ cell endodermal sinus tumour stage II Ovarian germ cell endodermal sinus tumour stage III Ovarian germ cell endodermal sinus tumour stage IV Ovarian germ cell polyembryoma Ovarian germ cell polyembryoma stage Ovarian germ cell polyembryoma stage Ovarian germ cell polyembryoma stage Ovarian germ cell polyembryoma stage Ovarian germ cell teratoma Ovarian germ cell teratoma stage I Ovarian germ cell teratoma stage II

## MedDRA v20.1 Preferred Term (PT)

Adult T-cell lymphoma/leukaemia stage Adult T-cell lymphoma/leukaemia stage Adult T-cell lymphoma/leukaemia stage Adult T-cell lymphoma/leukaemia stage Aesthesioneuroblastoma Alcoholisation procedure Aleukaemic leukaemia Alpha 1 foetoprotein abnormal Alpha 1 foetoprotein increased Alpha interferon therapy Alpha-L-fucosidase increased Alveolar rhabdomyosarcoma Alveolar soft part sarcoma Alveolar soft part sarcoma metastatic Alveolar soft part sarcoma recurrent Anal cancer Anal cancer metastatic Anal cancer recurrent Anal cancer stage 0 Anal cancer stage I Anal cancer stage II Anal cancer stage III Anal cancer stage IV Anal neoplasm Anal squamous cell carcinoma Anaplastic astrocytoma Anaplastic large cell lymphoma T- and

null-cell types refractory
Anaplastic large cell lymphoma T- and
null-cell types stage I
Anaplastic large cell lymphoma T- and
null-cell types stage II
Anaplastic large cell lymphoma T- and
null-cell types stage III
Anaplastic large cell lymphoma T- and
null-cell types stage IV
Anaplastic large-cell lymphoma
Anaplastic large-cell lymphoma
Anaplastic oligodendroglioma
Anaplastic oligodendroglioma
Anaplastic thyroid cancer
Androgen therapy
Angiocentric glioma

Anaplastic large cell lymphoma T- and

Anaplastic large cell lymphoma T- and

null-cell types

null-cell types recurrent

Angiocentric lymphoma

Angiocentric lymphoma recurrent

Angiocentric lymphoma refractory

Angiocentric lymphoma stage I

Angiocentric lymphoma stage II

Angiocentric lymphoma stage III

Histiocytic medullary reticulosis Histiocytic sarcoma Hodgkin's disease Hodgkin's disease lymphocyte depletion stage I site unspecified Hodgkin's disease lymphocyte depletion stage I subdiaphragm Hodgkin's disease lymphocyte depletion stage I supradiaphragm Hodgkin's disease lymphocyte depletion stage II site unspecified Hodgkin's disease lymphocyte depletion stage II subdiaphragm Hodgkin's disease lymphocyte depletion stage II supradiaphragm Hodgkin's disease lymphocyte depletion type recurrent Hodgkin's disease lymphocyte depletion type refractory Hodgkin's disease lymphocyte depletion type stage III Hodgkin's disease lymphocyte depletion type stage IV Hodgkin's disease lymphocyte depletion type stage unspecified Hodgkin's disease lymphocyte predominance stage I site unspec Hodgkin's disease lymphocyte predominance stage I subdiaphragm Hodgkin's disease lymphocyte predominance stage I supradiaphragm Hodgkin's disease lymphocyte predominance stage II site unspec Hodgkin's disease lymphocyte predominance stage II subdiaphragm Hodgkin's disease lymphocyte predominance stage II supradiaphragm Hodgkin's disease lymphocyte predominance type recurrent Hodgkin's disease lymphocyte predominance type refractory Hodgkin's disease lymphocyte predominance type stage III Hodgkin's disease lymphocyte predominance type stage IV Hodgkin's disease lymphocyte predominance type stage unspecified Hodgkin's disease mixed cellularity recurrent Hodgkin's disease mixed cellularity refractory Hodgkin's disease mixed cellularity stage I site unspecified Hodgkin's disease mixed cellularity

Ovarian germ cell teratoma stage III
Ovarian germ cell teratoma stage IV
Ovarian germ cell tumour
Ovarian germ cell tumour mixed
Ovarian granulosa cell tumour
Ovarian granulosa-theca cell tumour
Ovarian low malignant potential
tumour
Ovarian neoplasm
Ovarian Sertoli-Leydig cell tumour
Ovarian stromal cancer

Ovarian theca cell tumour

Paget's disease of nipple Paget's disease of penis Paget's disease of the vulva Palliative care Pancoast's tumour Pancreastatin abnormal Pancreastatin increased Pancreatectomy Pancreatic carcinoma Pancreatic carcinoma metastatic Pancreatic carcinoma recurrent Pancreatic carcinoma stage 0 Pancreatic carcinoma stage I Pancreatic carcinoma stage II Pancreatic carcinoma stage III Pancreatic carcinoma stage IV Pancreatic neoplasm Pancreatic neuroendocrine tumour Pancreatic neuroendocrine tumour metastatic Pancreatic sarcoma Pancreaticoduodenectomy Pancreaticosplenectomy Pancreatoblastoma Papillary renal cell carcinoma Papillary serous endometrial carcinoma Papillary thyroid cancer Paraganglion neoplasm Paraganglion neoplasm malignant Paranasal biopsy abnormal Paranasal sinus and nasal cavity malignant neoplasm Paranasal sinus and nasal cavity malignant neoplasm recurrent Paranasal sinus and nasal cavity malignant neoplasm stage 0 Paranasal sinus and nasal cavity malignant neoplasm stage I Paranasal sinus and nasal cavity malignant neoplasm stage II Paranasal sinus and nasal cavity

malignant neoplasm stage III

Paranasal sinus and nasal cavity

Hodgkin's disease mixed cellularity

stage I subdiaphragmatic

## MedDRA v20.1 Preferred Term (PT)

Angiocentric lymphoma stage IV Angiogenesis biomarker increased Angioimmunoblastic T-cell lymphoma Angioimmunoblastic T-cell lymphoma recurrent Angioimmunoblastic T-cell lymphoma refractory Angioimmunoblastic T-cell lymphoma stage I Angioimmunoblastic T-cell lymphoma stage II Angioimmunoblastic T-cell lymphoma stage III Angioimmunoblastic T-cell lymphoma stage IV Angiosarcoma Angiosarcoma metastatic Angiosarcoma non-metastatic Angiosarcoma recurrent Antiandrogen therapy Anti-NMDA antibody positive Antioestrogen therapy Anti-VGCC antibody positive Apocrine breast carcinoma Appendix cancer **APUDoma** Astroblastoma Astrocytoma Astrocytoma malignant Atypical fibroxanthoma Atypical teratoid/rhabdoid tumour of Autologous bone marrow transplantation therapy Axillary lymphadenectomy B precursor type acute leukaemia Basal cell carcinoma Basosquamous carcinoma Basosquamous carcinoma of skin B-cell depletion therapy B-cell lymphoma B-cell lymphoma recurrent B-cell lymphoma refractory B-cell lymphoma stage I B-cell lymphoma stage II B-cell lymphoma stage III B-cell lymphoma stage IV B-cell prolymphocytic leukaemia B-cell small lymphocytic lymphoma B-cell small lymphocytic lymphoma recurrent B-cell small lymphocytic lymphoma refractory B-cell small lymphocytic lymphoma

B-cell small lymphocytic lymphoma

stage I supradiaphragmatic Hodgkin's disease mixed cellularity stage II subdiaphragmatic Hodgkin's disease mixed cellularity stage II supradiaphragmatic Hodgkin's disease mixed cellularity stage III Hodgkin's disease mixed cellularity stage IV Hodgkin's disease mixed cellularity stage unspecified Hodgkin's disease nodular sclerosis Hodgkin's disease nodular sclerosis recurrent Hodgkin's disease nodular sclerosis refractory Hodgkin's disease nodular sclerosis Hodgkin's disease nodular sclerosis Hodgkin's disease nodular sclerosis stage III Hodgkin's disease nodular sclerosis stage IV Hodgkin's disease recurrent Hodgkin's disease refractory Hodgkin's disease stage I Hodgkin's disease stage II Hodgkin's disease stage III Hodgkin's disease stage IV Hodgkin's disease unclassifiable Hormone refractory breast cancer Hormone suppression therapy Hormone therapy Hormone-dependent prostate cancer Hormone-refractory prostate cancer Hormone-secreting ovarian tumour Huerthle cell carcinoma Human chorionic gonadotropin increased Human chorionic gonadotropin positive Human epidermal growth factor receptor increased Hypercalcaemia of malignancy Hyperleukocytosis Hyperthermia therapy Hypopharyngeal cancer Hypopharyngeal cancer recurrent Hypopharyngeal cancer stage 0 Hypopharyngeal cancer stage I Hypopharyngeal cancer stage II Hypopharyngeal cancer stage III Hypopharyngeal cancer stage IV Hypopharyngeal neoplasm Hypophysectomy

malignant neoplasm stage IV Paranasal sinus neoplasm Paraneoplastic arthritis Paraneoplastic dermatomyositis Paraneoplastic dermatosis Paraneoplastic encephalomyelitis Paraneoplastic glomerulonephritis Paraneoplastic nephrotic syndrome Paraneoplastic neurological syndrome Paraneoplastic pemphigus Paraneoplastic pleural effusion Paraneoplastic rash Paraneoplastic syndrome Parathyroid scan abnormal Parathyroid tumour Parathyroid tumour malignant Parathyroidectomy Parotidectomy Pelvic neoplasm Penile cancer Penile neoplasm Penile squamous cell carcinoma Penis carcinoma metastatic Penis carcinoma recurrent Penis carcinoma stage I Penis carcinoma stage II Penis carcinoma stage III Penis carcinoma stage IV Pepsinogen test positive Percutaneous ethanol injection therapy Pericardial effusion malignant Pericardial mesothelioma malignant Pericardial mesothelioma malignant recurrent Pericardial neoplasm Pericarditis malignant Peripheral nerve sheath tumour malignant Peripheral nervous system neoplasm Peripheral neuroepithelioma of bone Peripheral neuroepithelioma of bone metastatic Peripheral neuroepithelioma of bone recurrent Peripheral neuroepithelioma of soft Peripheral primitive neuroectodermal bone tumour Peripheral primitive neuroectodermal tumour of soft tissue Peripheral T-cell lymphoma unspecified Peripheral T-cell lymphoma unspecified recurrent Peripheral T-cell lymphoma unspecified refractory

## MedDRA v20.1 Preferred Term (PT)

stage II

B-cell small lymphocytic lymphoma stage III

B-cell small lymphocytic lymphoma

B-cell type acute leukaemia

B-cell unclassifiable lymphoma high

B-cell unclassifiable lymphoma low grade

Beta interferon therapy

Bile duct adenocarcinoma

Bile duct adenosquamous carcinoma

Bile duct cancer

Bile duct cancer recurrent

Bile duct cancer stage 0

Bile duct cancer stage I

Bile duct cancer stage II

Bile duct cancer stage III

Bile duct cancer stage IV

Bile duct squamous cell carcinoma

Biliary cancer metastatic

Biliary neoplasm

Biopsy abdominal wall abnormal

Biopsy adrenal gland abnormal

Biopsy anus abnormal

Biopsy artery abnormal

Biopsy bile duct abnormal

Biopsy bladder abnormal

Biopsy blood vessel abnormal

Biopsy bone abnormal

Biopsy bone marrow abnormal

Biopsy brain abnormal

Biopsy breast abnormal

Biopsy bronchus abnormal

Biopsy cartilage abnormal

Biopsy cervix abnormal

Biopsy chest wall abnormal

Biopsy chorionic villous abnormal

Biopsy colon abnormal

Biopsy conjunctiva abnormal

Biopsy cornea abnormal

Biopsy diaphragm abnormal

Biopsy ear abnormal

Biopsy endometrium abnormal

Biopsy epididymis abnormal

Biopsy eyelid abnormal

Biopsy fallopian tube abnormal

Biopsy foetal abnormal

Biopsy gallbladder abnormal

Biopsy heart abnormal

Biopsy intestine abnormal Biopsy kidney abnormal

Biopsy larynx abnormal

Biopsy ligament abnormal

Biopsy lip abnormal

Hysterectomy

Hysterosalpingectomy

Hysterosalpingo-oophorectomy

IDH differentiation syndrome

Ileectomy

Ileocolectomy Imaging procedure abnormal

Immune enhancement therapy

Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma

Immunoblastic lymphoma

Immunochemotherapy

In vivo gene therapy

Infected neoplasm

Inferior vena cava syndrome

Inflammatory carcinoma of breast

Inflammatory carcinoma of breast

stage III

Inflammatory carcinoma of breast

stage IV

Inflammatory carcinoma of the breast

Inflammatory malignant fibrous

histiocytoma

Inflammatory myofibroblastic tumour

Insulinoma

Interleukin therapy

Intestinal adenocarcinoma

Intestinal metastasis

Intestinal resection

Intestinal T-cell lymphoma recurrent

Intestinal T-cell lymphoma refractory Intestinal T-cell lymphoma stage I

Intestinal T-cell lymphoma stage II Intestinal T-cell lymphoma stage III

Intestinal T-cell lymphoma stage IV

Intracranial germ cell tumour

Intracranial meningioma malignant

Intracranial tumour haemorrhage Intraductal papillary breast neoplasm

Intraductal papillary-mucinous carcinoma of pancreas

Intraductal proliferative breast lesion

Intraocular melanoma

Intraperitoneal hyperthermic

chemotherapy

Intratumoural aneurysm Invasive breast carcinoma

Invasive ductal breast carcinoma

Invasive lobular breast carcinoma Invasive papillary breast carcinoma

Iris melanoma

Iris neoplasm

Jejunectomy Joint neoplasm

Juvenile chronic myelomonocytic

Peripheral T-cell lymphoma

unspecified stage I

Peripheral T-cell lymphoma

unspecified stage II

Peripheral T-cell lymphoma

unspecified stage III

Peripheral T-cell lymphoma

unspecified stage IV

Peritoneal carcinoma metastatic

Peritoneal fluid protein increased

Peritoneal mesothelioma malignant

Peritoneal mesothelioma malignant recurrent

Peritoneal neoplasm

Peritoneal sarcoma

Peritonectomy

Peritumoural oedema

Phaeochromocytoma

Phaeochromocytoma crisis

Phaeochromocytoma excision

Phaeochromocytoma malignant

Pharyngeal cancer

Pharyngeal cancer metastatic

Pharyngeal cancer recurrent

Pharyngeal cancer stage 0

Pharyngeal cancer stage I

Pharyngeal cancer stage II

Pharvngeal cancer stage III

Pharyngeal cancer stage IV

Pharyngeal neoplasm Pharyngectomy

Philadelphia chromosome positive

Photodynamic diagnostic procedure

Photon radiation therapy

Photon radiation therapy to bladder

Photon radiation therapy to blood

Photon radiation therapy to bone

Photon radiation therapy to brain

Photon radiation therapy to breast Photon radiation therapy to colon

Photon radiation therapy to ear, nose,

or throat

Photon radiation therapy to liver Photon radiation therapy to lung

Photon radiation therapy to pancreas

Photon radiation therapy to pleura

Photon radiation therapy to prostate

Photon radiation therapy to skin Photon radiation therapy to soft tissue

Photon radiation therapy to thyroid

Photon radiation therapy to uterus Phyllodes tumour

Pilomatrix carcinoma

Pineal germinoma

Pineal neoplasm Pineal parenchymal neoplasm

## MedDRA v20.1 Preferred Term (PT)

Biopsy liver abnormal Biopsy lung abnormal Biopsy lymph gland abnormal Biopsy mucosa abnormal Biopsy muscle abnormal Biopsy oesophagus abnormal Biopsy ovary abnormal Biopsy palate abnormal Biopsy pancreas abnormal Biopsy parathyroid gland abnormal Biopsy penis abnormal Biopsy pericardium abnormal Biopsy peripheral nerve abnormal Biopsy peritoneum abnormal Biopsy pharynx abnormal Biopsy pleura abnormal Biopsy prostate abnormal Biopsy rectum abnormal Biopsy retina abnormal Biopsy salivary gland abnormal Biopsy sclera abnormal Biopsy seminal vesicle abnormal Biopsy site unspecified abnormal Biopsy skin abnormal Biopsy small intestine abnormal Biopsy spinal cord abnormal Biopsy spleen abnormal Biopsy stomach abnormal Biopsy tendon abnormal Biopsy testes abnormal Biopsy thymus gland abnormal Biopsy thyroid gland abnormal Biopsy tongue abnormal Biopsy trachea abnormal Biopsy urethra abnormal Biopsy uterus abnormal Biopsy vagina abnormal Biopsy vocal cord abnormal Biopsy vulva abnormal Biotherapy Biphasic mesothelioma Bladder adenocarcinoma recurrent Bladder adenocarcinoma stage 0 Bladder adenocarcinoma stage I Bladder adenocarcinoma stage II Bladder adenocarcinoma stage III Bladder adenocarcinoma stage IV Bladder adenocarcinoma stage unspecified Bladder cancer Bladder cancer recurrent Bladder cancer stage 0, with cancer in Bladder cancer stage 0, without cancer Bladder cancer stage I, with cancer in

leukaemia Kaposi's sarcoma Kaposi's sarcoma AIDS related Kaposi's sarcoma classical type Keratinising squamous cell carcinoma of nasopharynx Keratoacanthoma Lacrimal duct neoplasm Langerhans' cell histiocytosis Langerhans cell sarcoma Large cell lung cancer Large cell lung cancer metastatic Large cell lung cancer recurrent Large cell lung cancer stage 0 Large cell lung cancer stage I Large cell lung cancer stage II Large cell lung cancer stage III Large cell lung cancer stage IV Large granular lymphocytosis Large intestinal polypectomy Laryngeal cancer Laryngeal cancer metastatic Laryngeal cancer recurrent Laryngeal cancer stage 0 Laryngeal cancer stage I Laryngeal cancer stage II Laryngeal cancer stage III Larvngeal cancer stage IV Laryngeal neoplasm Laryngeal squamous cell carcinoma Laryngopharyngectomy Laser brain ablation Leiomyosarcoma Leiomyosarcoma metastatic Leiomyosarcoma recurrent Lentigo maligna Lentigo maligna recurrent Lentigo maligna stage I Lentigo maligna stage II Lentigo maligna stage III Lentigo maligna stage IV Leptomeningeal myelomatosis Leukaemia Leukaemia basophilic Leukaemia cutis Leukaemia granulocytic Leukaemia in remission Leukaemia monocytic Leukaemia recurrent Leukaemic cardiac infiltration Leukaemic infiltration Leukaemic infiltration extramedullary Leukaemic infiltration gingiva Leukaemic infiltration hepatic Leukaemic infiltration ovary

malignant Pinealoblastoma Pinealoma Pituitary cancer metastatic Pituitary gland radiotherapy Pituitary neoplasm malignant recurrent Pituitary tumour Pituitary tumour recurrent Placental neoplasm Plasma cell leukaemia Plasma cell leukaemia in remission Plasma cell myeloma Plasma cell myeloma in remission Plasma cell myeloma recurrent Plasmablastic lymphoma Plasmacytoma Pleomorphic adenoma Pleomorphic liposarcoma Pleomorphic malignant fibrous histiocytoma Pleural mesothelioma Pleural mesothelioma malignant Pleural mesothelioma malignant recurrent Pleural neoplasm Pleural sarcoma Pleurectomy PML/RAR alpha expression Pneumonectomy POEMS syndrome Polyneuropathy in malignant disease Poorly differentiated thyroid carcinoma Porocarcinoma Portal vein embolisation Post breast therapy pain syndrome Post transplant lymphoproliferative disorder Postcricoid cancer Posterior fossa syndrome Precursor B-lymphoblastic lymphoma Precursor B-lymphoblastic lymphoma recurrent Precursor B-lymphoblastic lymphoma refractory Precursor B-lymphoblastic lymphoma Precursor B-lymphoblastic lymphoma stage II Precursor B-lymphoblastic lymphoma stage III Precursor B-lymphoblastic lymphoma stage IV Precursor T-lymphoblastic lymphoma/leukaemia Precursor T-lymphoblastic lymphoma/leukaemia recurrent

Leukaemic infiltration pulmonary

## MedDRA v20.1 Preferred Term (PT)

Bladder cancer stage I, without cancer in situ Bladder cancer stage II Bladder cancer stage III Bladder cancer stage IV Bladder neck resection Bladder neoplasm Bladder neoplasm surgery Bladder squamous cell carcinoma recurrent Bladder squamous cell carcinoma stage unspecified Bladder transitional cell carcinoma Bladder transitional cell carcinoma metastatic Bladder transitional cell carcinoma recurrent Bladder transitional cell carcinoma stage Bladder transitional cell carcinoma stage Bladder transitional cell carcinoma stage Bladder transitional cell carcinoma stage Bladder transitional cell carcinoma stage Blast cell crisis Blast crisis in myelogenous leukaemia Blastic plasmacytoid dendritic cell neoplasia Blood chromogranin A increased Bone cancer Bone cancer metastatic Bone giant cell tumour Bone giant cell tumour malignant Bone marrow infiltration Bone marrow leukaemic cell infiltration Bone marrow reticulin fibrosis Bone marrow tumour cell infiltration Bone neoplasm Bone sarcoma Bone scan abnormal Borderline mucinous tumour of ovary

Borderline ovarian tumour

Leukaemic infiltration renal Leukaemic lymphoma Leukaemic retinopathy Leukostasis syndrome Levdig cell tumour of the testis Linitis plastica Lip and/or oral cavity cancer Lip and/or oral cavity cancer recurrent Lip and/or oral cavity cancer stage 0 Lip and/or oral cavity cancer stage I Lip and/or oral cavity cancer stage II Lip and/or oral cavity cancer stage III Lip and/or oral cavity cancer stage IV Lip neoplasm Lip neoplasm malignant stage unspecified Lip squamous cell carcinoma Liposarcoma Liposarcoma metastatic Liposarcoma recurrent Liver ablation Liver carcinoma ruptured Liver scan abnormal Lobular breast carcinoma in situ Lung adenocarcinoma Lung adenocarcinoma recurrent Lung adenocarcinoma stage 0 Lung adenocarcinoma stage I Lung adenocarcinoma stage II Lung adenocarcinoma stage III Lung adenocarcinoma stage IV Lung cancer metastatic Lung carcinoma cell type unspecified recurrent Lung carcinoma cell type unspecified stage 0 Lung carcinoma cell type unspecified stage I Lung carcinoma cell type unspecified stage II Lung carcinoma cell type unspecified stage III Lung carcinoma cell type unspecified stage IV Lung infiltration malignant Lung lobectomy Lung neoplasm Lung neoplasm malignant Lung neoplasm surgery Lung squamous cell carcinoma metastatic Lung squamous cell carcinoma recurrent Lung squamous cell carcinoma stage 0 Lung squamous cell carcinoma stage I

Precursor T-lymphoblastic lymphoma/leukaemia refractory Precursor T-lymphoblastic lymphoma/leukaemia stage I Precursor T-lymphoblastic lymphoma/leukaemia stage II Precursor T-lymphoblastic lymphoma/leukaemia stage III Precursor T-lymphoblastic lymphoma/leukaemia stage IV Primary cardiac lymphoma Primary effusion lymphoma Primary gastrointestinal follicular lymphoma Primary mediastinal large B-cell lymphoma Primary mediastinal large B-cell lymphoma recurrent Primary mediastinal large B-cell lymphoma refractory Primary mediastinal large B-cell lymphoma stage I Primary mediastinal large B-cell lymphoma stage II Primary mediastinal large B-cell lymphoma stage III Primary mediastinal large B-cell lymphoma stage IV Primitive neuroectodermal tumour Primitive neuroectodermal tumour metastatic Proctectomy Proctocolectomy Progesterone receptor assay positive Prolactin-producing pituitary tumour Prolymphocytic leukaemia Prophylactic chemotherapy Prostate ablation Prostate cancer Prostate cancer metastatic Prostate cancer recurrent Prostate cancer stage 0 Prostate cancer stage I Prostate cancer stage II Prostate cancer stage III Prostate cancer stage IV Prostate cryoablation Prostate interstitial hyperthermia therapy Prostatectomy Prostatic specific antigen abnormal Prostatic specific antigen increased Pseudoachalasia Pseudomyxoma peritonei Pseudosarcoma

Pulmonary resection

Lung squamous cell carcinoma stage II

## MedDRA v20.1 Preferred Term (PT)

Borderline serous tumour of ovary

Bowen's disease

Brachytherapy

Brachytherapy to eye

Brachytherapy to penis

Brachytherapy to tongue

Brachytherapy to tonsil

Brain cancer metastatic

Brain neoplasm

Brain neoplasm malignant

Brain sarcoma

Brain scan abnormal

Brain stem glioma

Brain teratoma

Brain tumour operation

Breast angiosarcoma

Breast angiosarcoma metastatic

Breast cancer

Breast cancer female

Breast cancer in situ

Breast cancer male

Breast cancer metastatic

Breast cancer recurrent

Breast cancer stage I

Breast cancer stage II

Breast cancer stage III

Breast cancer stage IV

Breast capsulotomy

Breast conserving surgery

Breast neoplasm

Breast prosthesis implantation

Breast reconstruction

Breast sarcoma

Breast sarcoma metastatic

Breast sarcoma recurrent

Breast tumour excision

Brenner tumour

Bronchial carcinoma

Bronchial neoplasm

Bronchioloalveolar carcinoma Burkitt's leukaemia

Burkitt's lymphoma

Burkitt's lymphoma recurrent Burkitt's lymphoma refractory

Burkitt's lymphoma stage I

Burkitt's lymphoma stage II

Burkitt's lymphoma stage III

Burkitt's lymphoma stage IV

Buschke-Lowenstein's tumour

Cancer hormonal therapy

Cancer in remission

Cancer pain

Cancer staging

Cancer surgery

Carbohydrate antigen 125 increased

Carbohydrate antigen 15-3 increased

Lung squamous cell carcinoma stage

Lung squamous cell carcinoma stage

Lymph nodes scan abnormal

Lymphadenectomy

Lymphangiosarcoma

Lymphangiosis carcinomatosa

Lymphatic mapping

Lymphatic system neoplasm

Lymphocyte adoptive therapy

Lymphocytic leukaemia

Lymphocytic lymphoma

Lymphoid leukaemia (in remission)

Lymphoma

Lymphoma AIDS related

Lymphoma cutis

Lymphoma operation

Lymphoma transformation

Lymphoplasmacytoid

lymphoma/immunocytoma

Lymphoplasmacytoid

lymphoma/immunocytoma recurrent

Lymphoplasmacytoid

lymphoma/immunocytoma refractory

Lymphoplasmacytoid

lymphoma/immunocytoma stage I

Lymphoplasmacytoid

lymphoma/immunocytoma stage II

Lymphoplasmacytoid

lymphoma/immunocytoma stage III

Lymphoplasmacytoid

lymphoma/immunocytoma stage IV

Lymphoproliferative disorder

Lymphoproliferative disorder in

remission

Male reproductive tract neoplasm

Malignant anorectal neoplasm

Malignant ascites

Malignant blue naevus

Malignant bowel obstruction

Malignant connective tissue neoplasm

Malignant cranial nerve neoplasm

Malignant dysphagia

Malignant exophthalmos

Malignant fibrous histiocytoma

Malignant fibrous histiocytoma

metastatic

Malignant fibrous histiocytoma of

bone

Malignant fibrous histiocytoma

recurrent

Malignant genitourinary tract

neoplasm

Malignant giant cell fibrous

histiocytoma

Pulmonary tumour thrombotic

microangiopathy

Pylorectomy

Pvoderma gangrenosum

Quevrat erythroplasia

Radiation therapy to ear, nose, or throat

Radical cystectomy

Radical hysterectomy

Radical mastectomy

Radical neck dissection

Radical prostatectomy

Radioactive iodine therapy

Radioembolisation

Radioisotope scan abnormal

Radiosensitisation therapy

Radiotherapy

Radiotherapy to abdomen

Radiotherapy to adrenal gland

Radiotherapy to blood

Radiotherapy to bone

Radiotherapy to brain

Radiotherapy to breast

Radiotherapy to colon Radiotherapy to ear

Radiotherapy to eye

Radiotherapy to gallbladder

Radiotherapy to gastrointestinal tract Radiotherapy to head and neck

Radiotherapy to joint

Radiotherapy to kidney

Radiotherapy to liver

Radiotherapy to lung

Radiotherapy to lymph nodes

Radiotherapy to mediastinum

Radiotherapy to nose

Radiotherapy to oesophagus

Radiotherapy to oral cavity Radiotherapy to ovary

Radiotherapy to pancreas

Radiotherapy to pleura

Radiotherapy to prostate

Radiotherapy to rectum

Radiotherapy to skin Radiotherapy to soft tissue

Radiotherapy to spleen

Radiotherapy to stomach

Radiotherapy to throat

Radiotherapy to thymus

Radiotherapy to thyroid Radiotherapy to urinary bladder

Radiotherapy to uterus

Radiotherapy to vagina Rectal adenocarcinoma

Rectal cancer

Rectal cancer metastatic Rectal cancer recurrent

## MedDRA v20.1 Preferred Term (PT)

Carbohydrate antigen 19-9 increased Carbohydrate antigen 27.29 increased Carbohydrate antigen 549 increased Carcinoembryonic antigen decreased Carcinoembryonic antigen increased Carcinoid crisis Carcinoid heart disease Carcinoid syndrome Carcinoid tumour Carcinoid tumour of the appendix Carcinoid tumour of the caecum Carcinoid tumour of the duodenum Carcinoid tumour of the gastrointestinal tract Carcinoid tumour of the pancreas Carcinoid tumour of the prostate Carcinoid tumour of the small bowel Carcinoid tumour of the stomach Carcinoid tumour pulmonary Carcinoma ex-pleomorphic adenoma Carcinoma in situ Carcinoma in situ of eye Carcinoma in situ of penis Carcinoma in situ of skin Carcinoma in situ of trachea Carcinomatous polyarthritis Cardiac neoplasm malignant Cardiac neoplasm unspecified Cardiac teratoma Carotid body tumour Cartilage neoplasm CD20 antigen positive CD25 antigen positive CD30 expression Cell marker increased Cell-free and concentrated ascites reinfusion therapy Cementoplasty Central nervous system leukaemia Central nervous system lymphoma Central nervous system melanoma Central nervous system neoplasm Central nervous system neuroblastoma Cerebellar tumour Cerebellopontine angle tumour Cervical tumour excision Cervix cancer metastatic Cervix carcinoma Cervix carcinoma recurrent Cervix carcinoma stage 0 Cervix carcinoma stage I Cervix carcinoma stage II Cervix carcinoma stage III Cervix carcinoma stage IV

Cervix neoplasm

Chemotherapy

Malignant glioma Malignant haemangiopericytoma Malignant haemangiopericytoma metastatic Malignant haemangiopericytoma recurrent Malignant histiocytosis Malignant hydatidiform mole Malignant joint neoplasm Malignant lymphoid neoplasm Malignant lymphoma unclassifiable high grade Malignant lymphoma unclassifiable low grade Malignant mast cell neoplasm Malignant mediastinal neoplasm Malignant melanoma Malignant melanoma in situ Malignant melanoma of evelid Malignant melanoma of sites other than skin Malignant melanoma stage I Malignant melanoma stage II Malignant melanoma stage III Malignant melanoma stage IV Malignant meningioma metastatic Malignant mesenchymoma Malignant mesenchymoma metastatic Malignant mesenchymoma recurrent Malignant mesenteric neoplasm Malignant middle ear neoplasm Malignant muscle neoplasm Malignant neoplasm of ampulla of Vater Malignant neoplasm of auricular cartilage Malignant neoplasm of choroid Malignant neoplasm of conjunctiva Malignant neoplasm of cornea Malignant neoplasm of eye Malignant neoplasm of eyelid Malignant neoplasm of islets of Langerhans Malignant neoplasm of lacrimal duct Malignant neoplasm of lacrimal gland Malignant neoplasm of orbit Malignant neoplasm of paraurethral glands Malignant neoplasm of placenta Malignant neoplasm of pleura Malignant neoplasm of pleura metastatic Malignant neoplasm of renal pelvis Malignant neoplasm of retina Malignant neoplasm of seminal vesicle Malignant neoplasm of spermatic cord

Rectal cancer stage 0 Rectal cancer stage I Rectal cancer stage II Rectal cancer stage III Rectal cancer stage IV Rectal neoplasm Rectosigmoid cancer Rectosigmoid cancer metastatic Rectosigmoid cancer recurrent Rectosigmoid cancer stage 0 Rectosigmoid cancer stage I Rectosigmoid cancer stage II Rectosigmoid cancer stage III Rectosigmoid cancer stage IV Recurrent cancer Refractory cancer Regional chemotherapy Renal cancer Renal cancer metastatic Renal cancer recurrent Renal cancer stage I Renal cancer stage II Renal cancer stage III Renal cancer stage IV Renal cell carcinoma Renal cell carcinoma recurrent Renal cell carcinoma stage I Renal cell carcinoma stage II Renal cell carcinoma stage III Renal cell carcinoma stage IV Renal neoplasm Renal scan abnormal Renal tumour excision Respiratory tract carcinoma in situ Respiratory tract neoplasm Retinal melanoma Retinal neoplasm Retinal tumour excision Retinoblastoma Retro-orbital neoplasm Retroperitoneal cancer Retroperitoneal neoplasm Retroperitoneal neoplasm metastatic Retro-pubic prostatectomy Rhabdoid tumour Rhabdoid tumour of the kidney Rhabdomyosarcoma Rhabdomyosarcoma recurrent Richter's syndrome Round cell liposarcoma Salivary bypass tube insertion Salivary gland cancer Salivary gland cancer recurrent Salivary gland cancer stage 0 Salivary gland cancer stage I

Salivary gland cancer stage II

## MedDRA v20.1 Preferred Term (PT)

Chemotherapy cardiotoxicity attenuation Chemotherapy cytokine prophylaxis Chemotherapy extravasation

management

Chemotherapy multiple agents systemic Chemotherapy neurotoxicity attenuation Chemotherapy sensitivity and resistance

Chemotherapy single agent systemic Chemotherapy urothelial toxicity

attenuation

Chest wall tumour

Chloroma

Chloroma (in remission) Cholangiocarcinoma Cholangiosarcoma

Chondrosarcoma

Chondrosarcoma metastatic Chondrosarcoma recurrent

Chordoma

Choriocarcinoma Choroid melanoma Choroid neoplasm

Choroid plexus carcinoma Choroid tumour excision

Chronic eosinophilic leukaemia

Chronic leukaemia

Chronic leukaemia in remission Chronic lymphocytic leukaemia Chronic lymphocytic leukaemia (in remission)

Chronic lymphocytic leukaemia recurrent

Cl : 1

Chronic lymphocytic leukaemia refractory

Chronic lymphocytic leukaemia stage 0 Chronic lymphocytic leukaemia stage 1 Chronic lymphocytic leukaemia stage 2 Chronic lymphocytic leukaemia stage 3 Chronic lymphocytic leukaemia stage 4

Chronic lymphocytic leukaemia

transformation

Chronic myeloid leukaemia (in remission)

Chronic myeloid leukaemia recurrent Chronic myeloid leukaemia

transformation

Chronic myelomonocytic leukaemia Chronic myelomonocytic leukaemia (in

remission)

C-kit gene negative
Clear cell carcinoma of cervix
Clear cell endometrial carcinoma
Clear cell renal cell carcinoma
Clear cell sarcoma of soft tissue

Malignant neoplasm of spinal cord Malignant neoplasm of thorax Malignant neoplasm of thymus Malignant neoplasm of unknown primary site

Malignant neoplasm of uterine adnexa Malignant neoplasm papilla of Vater Malignant neoplasm progression Malignant nervous system neoplasm

Malignant nipple neoplasm
Malignant nipple neoplasm female

Malignant nipple neoplasm male Malignant oligodendroglioma

Malignant ovarian cyst Malignant palate neoplasm

Malignant pericardial neoplasm Malignant peritoneal neoplasm

Malignant pituitary tumour Malignant pleural effusion

Malignant polyp

Malignant psoas syndrome

Malignant respiratory tract neoplasm

Malignant splenic neoplasm Malignant sweat gland neoplasm Malignant transformation

Malignant urinary tract neoplasm

Mantle cell lymphoma

Mantle cell lymphoma recurrent Mantle cell lymphoma refractory Mantle cell lymphoma stage I

Mantle cell lymphoma stage I Mantle cell lymphoma stage II Mantle cell lymphoma stage IV

Marginal zone lymphoma

Marginal zone lymphoma recurrent Marginal zone lymphoma refractory Marginal zone lymphoma stage I Marginal zone lymphoma stage II

Marginal zone lymphoma stage III Marginal zone lymphoma stage IV

Marjolin's ulcer Mastectomy

Mastocytic leukaemia

Mastoidectomy

Maternal cancer in pregnancy Mature B-cell type acute leukaemia Maxillofacial sinus neoplasm

Mediastinal biopsy abnormal Mediastinum neoplasm

Medullary carcinoma of breast Medullary thyroid cancer

Medulloblastoma

Medulloblastoma recurrent

Meigs' syndrome Melanoma recurrent Meningeal neoplasm Salivary gland cancer stage III Salivary gland cancer stage IV

Salivary gland neoplasm

Salivary gland resection Salivary gland scan abnormal

Salpingectomy

Salpingo-oophorectomy

Salpingo-oophorectomy bilateral Salpingo-oophorectomy unilateral

Sarcoma

Sarcoma excision
Sarcoma metastatic
Sarcoma of skin
Sarcoma uterus

Sarcomatoid mesothelioma

Sarcomatosis

Scan abdomen abnormal

Scan abnormal

Scan adrenal gland abnormal Scan bone marrow abnormal Scan gallium abnormal

Scan myocardial perfusion abnormal

Scan with contrast abnormal

Scrotal cancer

Sebaceous carcinoma Second primary malignancy

Secondary cerebellar degeneration

Secretory adenoma of pituitary

Seminoma

Serous cystadenocarcinoma of pancreas

pancreas

Serous cystadenocarcinoma ovary Sertoli cell testicular tumour

Sigmoidectomy

Signet-ring cell carcinoma Simple mastectomy Sinus cancer metastatic Skin angiosarcoma

Skin cancer

Skin cancer metastatic Skin cryotherapy

Skin neoplasm bleeding Skin neoplasm bleeding Skin neoplasm excision

Skin squamous cell carcinoma metastatic

Small cell carcinoma

Small cell carcinoma of the cervix

Small cell lung cancer

Small intestine carcinoma

Small cell lung cancer extensive stage
Small cell lung cancer limited stage
Small cell lung cancer metastatic
Small cell lung cancer recurrent
Small intestinal resection
Small intestine adenocarcinoma

## MedDRA v20.1 Preferred Term (PT)

Clear cell sarcoma of the kidney Clonal evolution CNS germinoma

Colectomy Colectomy total

Colon cancer

Colon cancer metastatic Colon cancer recurrent Colon cancer stage 0

Colon cancer stage I

Colon cancer stage II Colon cancer stage III

Colon cancer stage IV

Colon neoplasm

Colony stimulating factor therapy

Colorectal adenocarcinoma

Colorectal cancer

Colorectal cancer metastatic Colorectal cancer recurrent Colorectal cancer stage I

Colorectal cancer stage II

Colorectal cancer stage III Colorectal cancer stage IV Colorectal carcinoma stage 0

Composite lymphoma

Computerised tomogram breast

abnormal

Computerised tomogram liver abnormal

Congenital fibrosarcoma

Congenital malignant neoplasm Congenital neoplasm

Congenital retinoblastoma Congenital teratoma Conjunctival melanoma

Conjunctival neoplasm Conjunctival primary acquired

melanosis

Connective tissue neoplasm Cutaneous lymphoma

Cyclotron therapy

Cystadenocarcinoma ovary

Cystoprostatectomy Cytokeratin 18 increased

Dedifferentiated liposarcoma Dermatofibrosarcoma protuberans

Dermatofibrosarcoma protuberans

metastatic

Desmoplastic melanoma Desmoplastic mesothelioma

Desmoplastic small round cell tumour

Diaphragm neoplasm

Diffuse large B-cell lymphoma

Diffuse large B-cell lymphoma recurrent

Diffuse large B-cell lymphoma

refractory

Diffuse large B-cell lymphoma stage I

Meningioma malignant

Mesenteric neoplasm

Mesothelioma

Mesothelioma malignant

Mesothelioma malignant recurrent

Metaplastic breast carcinoma Metastases to abdominal cavity

Metastases to abdominal wall

Metastases to adrenals

Metastases to biliary tract Metastases to bladder

Metastases to bone

Metastases to bone marrow

Metastases to breast

Metastases to central nervous system

Metastases to chest wall Metastases to diaphragm

Metastases to Eustachian tube

Metastases to eve

Metastases to fallopian tube Metastases to gallbladder

Metastases to gastrointestinal tract

Metastases to heart Metastases to kidney

Metastases to larynx

Metastases to liver Metastases to lung

Metastases to lymph nodes

Metastases to meninges Metastases to mouth

Metastases to muscle Metastases to nasal sinuses

Metastases to neck

Metastases to nervous system Metastases to oesophagus

Metastases to ovary Metastases to pancreas

Metastases to pelvis Metastases to penis

Metastases to perineum Metastases to peripheral nervous

system

Metastases to peripheral vascular

system

Metastases to peritoneum

Metastases to pharynx Metastases to pituitary gland

Metastases to placenta Metastases to pleura

Metastases to prostate Metastases to rectum

Metastases to reproductive organ Metastases to retroperitoneum

Metastases to skin Metastases to soft tissue

Metastases to salivary gland

Small intestine carcinoma metastatic

Small intestine carcinoma recurrent

Small intestine carcinoma stage 0

Small intestine carcinoma stage I

Small intestine carcinoma stage II

Small intestine carcinoma stage III

Small intestine carcinoma stage IV Small intestine leiomyosarcoma

Smooth muscle cell neoplasm

Soft tissue neoplasm

Soft tissue sarcoma

Solid pseudopapillary tumour of the pancreas

Somatostatin receptor scan abnormal

Somatostatinoma

Spermatocytic seminoma Spinal cord neoplasm

Spinal meningioma malignant

Spindle cell sarcoma Spleen scan abnormal

Splenectomy

Splenic marginal zone lymphoma

Splenic marginal zone lymphoma

recurrent

Splenic marginal zone lymphoma

refractory

Splenic marginal zone lymphoma stage

Splenic marginal zone lymphoma stage

Splenic marginal zone lymphoma stage

Splenic marginal zone lymphoma stage

Splenic neoplasm malignancy

unspecified

Squamous cell breast carcinoma

Squamous cell carcinoma

Squamous cell carcinoma of head and

neck

Squamous cell carcinoma of lung Squamous cell carcinoma of pharynx

Squamous cell carcinoma of skin Squamous cell carcinoma of the cervix

Squamous cell carcinoma of the

hypopharynx Squamous cell carcinoma of the oral

cavity Squamous cell carcinoma of the tongue Squamous cell carcinoma of the vagina Squamous cell carcinoma of the vulva

Squamous endometrial carcinoma Stauffer's syndrome Stem cell transplant Stewart-Treves syndrome Stomach scan abnormal

## MedDRA v20.1 Preferred Term (PT)

Diffuse large B-cell lymphoma stage II Diffuse large B-cell lymphoma stage III Diffuse large B-cell lymphoma stage IV Diffuse uveal melanocytic proliferation Disseminated large cell lymphoma Double hit lymphoma Ductal adenocarcinoma of pancreas Duodenal neoplasm Duodenectomy Dysplastic naevus syndrome Ear neoplasm Ear neoplasm malignant Eastern Cooperative Oncology Group performance status improved Eastern Cooperative Oncology Group performance status worsened Eccrine carcinoma Ectopic ACTH syndrome Ectopic aldosterone secretion Ectopic antidiuretic hormone secretion Ectopic calcitonin production Ectopic chorionic gonadotrophin secretion Ectopic growth hormone secretion Ectopic hormone secretion Ectopic parathyroid hormone production Ectopic prolactin secretion Ectopic renin secretion Electron radiation therapy Electron radiation therapy to bladder Electron radiation therapy to blood Electron radiation therapy to bone Electron radiation therapy to brain Electron radiation therapy to breast Electron radiation therapy to colon Electron radiation therapy to ear, nose, or throat Electron radiation therapy to liver Electron radiation therapy to lung Electron radiation therapy to pancreas Electron radiation therapy to prostate Electron radiation therapy to skin Electron radiation therapy to soft tissue Electron radiation therapy to uterus Elephantiasis nostras verrucosa Embryonal rhabdomyosarcoma Endocrine neoplasm Endocrine neoplasm malignant Endometrial adenocarcinoma Endometrial cancer Endometrial cancer metastatic Endometrial cancer recurrent Endometrial cancer stage 0 Endometrial cancer stage I Endometrial cancer stage II

Endometrial cancer stage III

Metastases to spinal cord Metastases to spine Metastases to spleen Metastases to stomach Metastases to testicle Metastases to the mediastinum Metastases to the respiratory system Metastases to thorax Metastases to thyroid Metastases to tonsils Metastases to trachea Metastases to urinary tract Metastases to uterus Metastases to vagina Metastasis Metastatic bronchial carcinoma Metastatic carcinoid tumour Metastatic carcinoma of the bladder Metastatic choriocarcinoma Metastatic gastric cancer Metastatic glioma Metastatic glucagonoma Metastatic lymphoma Metastatic malignant melanoma Metastatic neoplasm Metastatic nervous system neoplasm Metastatic ocular melanoma Metastatic pulmonary embolism Metastatic renal cell carcinoma Metastatic salivary gland cancer Metastatic squamous cell carcinoma Metastatic uterine cancer Microsatellite instability cancer Minimal residual disease Mismatch repair cancer syndrome Mixed adenoneuroendocrine carcinoma Mixed hepatocellular cholangiocarcinoma Mixed-type liposarcoma Modified radical mastectomy Monoclonal gammopathy Monocytic leukaemia in remission Mucinous adenocarcinoma of appendix Mucinous breast carcinoma Mucinous cystadenocarcinoma of pancreas Mucinous cystadenocarcinoma ovary Mucinous endometrial carcinoma Mucoepidermoid carcinoma Mucoepidermoid carcinoma of salivary gland Mueller's mixed tumour Multiple gated acquisition scan

Superficial spreading melanoma stage I Superficial spreading melanoma stage Superficial spreading melanoma stage Superficial spreading melanoma stage Superficial spreading melanoma stage unspecified Superior vena cava occlusion Superior vena cava syndrome Suprapubic prostatectomy Synovial sarcoma Synovial sarcoma metastatic Synovial sarcoma recurrent Targeted cancer therapy T-cell chronic lymphocytic leukaemia T-cell lymphoma T-cell lymphoma recurrent T-cell lymphoma refractory T-cell lymphoma stage I T-cell lymphoma stage II T-cell lymphoma stage III T-cell lymphoma stage IV T-cell prolymphocytic leukaemia T-cell type acute leukaemia T-cell unclassifiable lymphoma high grade T-cell unclassifiable lymphoma low grade Tendon neoplasm Teratoma Testicular cancer metastatic Testicular choriocarcinoma Testicular choriocarcinoma recurrent Testicular choriocarcinoma stage I Testicular choriocarcinoma stage II Testicular choriocarcinoma stage III Testicular embryonal carcinoma Testicular embryonal carcinoma stage I Testicular embryonal carcinoma stage Testicular embryonal carcinoma stage Testicular germ cell cancer Testicular germ cell cancer metastatic Testicular germ cell tumour Testicular germ cell tumour mixed Testicular germ cell tumour mixed stage I Testicular germ cell tumour mixed stage II Testicular germ cell tumour mixed stage III Testicular leiomyosarcoma Testicular malignant teratoma

abnormal

## MedDRA v20.1 Preferred Term (PT)

Endometrial cancer stage IV Endometrial neoplasm Endometrial sarcoma Endometrial sarcoma metastatic Endometrial sarcoma recurrent Endometrial stromal sarcoma

Endotheliomatosis

Enteropathy-associated T-cell

lymphoma

Eosinophilic leukaemia

Ependymoma Ependymoma malignant Epididymal cancer Epididymal neoplasm Epiglottic carcinoma Epiglottidectomy Epithelioid mesothelioma Epithelioid sarcoma

Epithelioid sarcoma metastatic Epithelioid sarcoma recurrent Epstein Barr virus positive mucocutaneous ulcer

Epstein-Barr virus associated lymphoma

Epstein-Barr virus associated lymphoproliferative disorder

Erythraemic myelosis (in remission)

Erythroleukaemia Ewing's sarcoma

Ewing's sarcoma metastatic Ewing's sarcoma recurrent Ex vivo gene therapy Exploratory operation

Extended radical mastectomy Extradural neoplasm

Extragonadal primary embryonal

carcinoma

Extragonadal primary germ cell tumour Extragonadal primary germ cell tumour mixed

Extragonadal primary germ cell tumour mixed stage I

Extragonadal primary germ cell tumour mixed stage II

Extragonadal primary germ cell tumour mixed stage III

Extragonadal primary malignant

teratoma

Extragonadal primary non-seminoma Extragonadal primary non-seminoma stage I

Extragonadal primary non-seminoma stage II

Extragonadal primary non-seminoma

stage III

Extragonadal primary non-seminoma stage IV

Muscle neoplasm

Musculoskeletal cancer Myasthenic syndrome Mycosis fungoides

Mycosis fungoides recurrent Mycosis fungoides refractory Mycosis fungoides stage I Mycosis fungoides stage II Mycosis fungoides stage III

Mycosis fungoides stage IV Myectomy Myeloblastoma Mveloid leukaemia

Myeloid leukaemia in remission

Myeloid metaplasia

Myeloma cast nephropathy Myeloproliferative neoplasm

Mvxofibrosarcoma Myxoid liposarcoma Naevoid melanoma Nasal cavity cancer Nasal neoplasm Nasal sinus cancer Nasopharyngeal cancer

Nasopharyngeal cancer metastatic Nasopharyngeal cancer recurrent Nasopharyngeal cancer stage 0 Nasopharvngeal cancer stage I Nasopharyngeal cancer stage II Nasopharyngeal cancer stage III Nasopharyngeal cancer stage IV Natural killer-cell leukaemia

Natural killer-cell lymphoblastic

lymphoma

Necrolytic migratory erythema Needle biopsy site unspecified

abnormal

Neoadjuvant therapy Neobladder surgery Neonatal leukaemia Neonatal neuroblastoma

Neoplasm

Neoplasm malignant Neoplasm of appendix

Neoplasm of cornea unspecified

malignancy Neoplasm of orbit Neoplasm of thymus Neoplasm progression Neoplasm prostate Neoplasm recurrence Neoplasm skin Neoplasm swelling Nephrectomy Nephroblastoma

Nephroureterectomy

Testicular malignant teratoma stage I Testicular malignant teratoma stage II

Testicular malignant teratoma stage III

Testicular neoplasm Testicular scan abnormal Testicular seminoma (pure)

Testicular seminoma (pure) stage I Testicular seminoma (pure) stage II Testicular seminoma (pure) stage III

Testicular yolk sac tumour

Testicular yolk sac tumour stage I Testicular yolk sac tumour stage II Testicular yolk sac tumour stage III

Testis cancer

Testis cancer recurrent

Throat cancer

Thymic cancer metastatic

Thymoma

Thymoma malignant

Thymoma malignant recurrent Thyroid B-cell lymphoma

Thyroid cancer

Thyroid cancer metastatic Thyroid cancer recurrent Thyroid cancer stage 0 Thyroid cancer stage I Thyroid cancer stage II Thyroid cancer stage III Thyroid cancer stage IV

Thyroid electron radiation therapy Thyroid gland scan abnormal

Thyroid neoplasm

Thyroid stimulating hormoneproducing pituitary tumour

Thyroidectomy

Tissue polypeptide antigen increased

Tongue cancer metastatic Tongue cancer recurrent Tongue carcinoma stage 0 Tongue carcinoma stage I Tongue carcinoma stage II Tongue carcinoma stage III Tongue carcinoma stage IV Tongue neoplasm

Tongue neoplasm malignant stage

unspecified Tonsil cancer Tonsil cancer metastatic Tonsillar neoplasm Total adrenalectomy Tracheal cancer Tracheal neoplasm Tracheal resection Transcatheter arterial

chemoembolisation

Transcranial electrical motor evoked

## MedDRA v20.1 Preferred Term (PT)

Extragonadal primary seminoma (pure) Extragonadal primary seminoma (pure) stage I

Extragonadal primary seminoma (pure) stage II

Extragonadal primary seminoma (pure) stage III

Extragonadal primary seminoma (pure) stage IV

Extramammary Paget's disease Extranodal marginal zone B-cell lymphoma (MALT type) Extranodal marginal zone B-cell lymphoma (MALT type) recurrent Extranodal marginal zone B-cell lymphoma (MALT type) refractory Extranodal marginal zone B-cell lymphoma (MALT type) stage I Extranodal marginal zone B-cell lymphoma (MALT type) stage II Extranodal marginal zone B-cell lymphoma (MALT type) stage III Extranodal marginal zone B-cell lymphoma (MALT type) stage IV Extraocular retinoblastoma Extra-osseous Ewing's sarcoma Extra-osseous Ewing's sarcoma

metastatic Extra-osseous Ewing's sarcoma recurrent

Extraskeletal chondrosarcoma metastatic Extraskeletal chondrosarcoma recurrent Extraskeletal myxoid chondrosarcoma

Extraskeletal osteosarcoma Extraskeletal osteosarcoma metastatic Extraskeletal osteosarcoma recurrent

Eyelid tumour

Fallopian tube cancer

Fallopian tube cancer metastatic Fallopian tube cancer stage I Fallopian tube cancer stage II Fallopian tube cancer stage III Fallopian tube cancer stage IV Fallopian tube neoplasm Familial medullary thyroid cancer

Female reproductive neoplasm

Female reproductive tract carcinoma in situ

Fibrosarcoma

Fibrosarcoma excision Fibrosarcoma metastatic Fiducial marker placement Fms-like tyrosine kinase 3 positive Follicle centre lymphoma diffuse small

cell lymphoma

Follicle centre lymphoma diffuse small

Nervous system neoplasm

Nervous system neoplasm surgery

Neuroblastoma

Neuroblastoma recurrent

Neuroectodermal neoplasm

Neuroendocrine breast tumour

Neuroendocrine carcinoma

Neuroendocrine carcinoma metastatic Neuroendocrine carcinoma of the

bladder

Neuroendocrine carcinoma of the skin

Neuroendocrine tumour

Neuroendocrine tumour of the lung Neuroendocrine tumour of the lung

metastatic Neuroendoscopy

Neurofibrosarcoma

Neurofibrosarcoma metastatic

Neurofibrosarcoma recurrent

Neuromyotonia

Neurotensinoma

Nipple neoplasm

Nipple resection

NMP22 test abnormal

Nodal marginal zone B-cell lymphoma Nodal marginal zone B-cell lymphoma recurrent

Nodal marginal zone B-cell lymphoma refractory

Nodal marginal zone B-cell lymphoma

Nodal marginal zone B-cell lymphoma

Nodal marginal zone B-cell lymphoma stage III

Nodal marginal zone B-cell lymphoma stage IV

Nodular lymphocyte predominant Hodgkin lymphoma

Nodular melanoma

Nongerminomatous germ cell tumour

of the CNS

Non-Hodgkin's lymphoma

Non-Hodgkin's lymphoma metastatic Non-Hodgkin's lymphoma recurrent

Non-Hodgkin's lymphoma refractory

Non-Hodgkin's lymphoma stage I Non-Hodgkin's lymphoma stage II

Non-Hodgkin's lymphoma stage III Non-Hodgkin's lymphoma stage IV

Non-Hodgkin's lymphoma transformed recurrent

Non-Hodgkin's lymphoma unspecified histology aggressive

Non-Hodgkin's lymphoma unspecified histology aggressive recurrent

potential monitoring abnormal Transformation to acute myeloid

leukaemia

Transitional cell cancer of renal pelvis

and ureter metastatic

Transitional cell cancer of the renal pelvis and ureter

Transitional cell cancer of the renal pelvis and ureter localised

Transitional cell cancer of the renal

pelvis and ureter recurrent

Transitional cell cancer of the renal pelvis and ureter regional

Transitional cell carcinoma

Transitional cell carcinoma metastatic

Transitional cell carcinoma recurrent

Transitional cell carcinoma urethra

Transurethral bladder resection

Transurethral prostatectomy

Triple hit lymphoma

Triple negative breast cancer

Trousseau's syndrome

Tubular breast carcinoma

Tumour associated fever

Tumour budding

Tumour cavitation

Tumour cell mobilisation

Tumour compression

Tumour embolism

Tumour excision

Tumour exudation

Tumour fistulisation

Tumour flare

Tumour haemorrhage

Tumour inflammation

Tumour invasion

Tumour lysis syndrome

Tumour marker abnormal

Tumour marker decreased Tumour marker increased

Tumour necrosis

Tumour obstruction

Tumour of ampulla of Vater

Tumour pain

Tumour perforation

Tumour pruritus

Tumour pseudoprogression

Tumour rupture

Tumour thrombosis

Tumour treating fields therapy

Tumour ulceration

Tumour vaccine therapy

Ultrasound pancreas abnormal

Ultrasound scan abnormal Ultrasound scan vagina abnormal

Undifferentiated carcinoma of colon

## MedDRA v20.1 Preferred Term (PT)

cell lymphoma recurrent Follicle centre lymphoma diffuse small cell lymphoma refractory Follicle centre lymphoma diffuse small cell lymphoma stage I Follicle centre lymphoma diffuse small cell lymphoma stage II Follicle centre lymphoma diffuse small cell lymphoma stage III Follicle centre lymphoma diffuse small cell lymphoma stage IV Follicle centre lymphoma, follicular grade I. II. III Follicle centre lymphoma, follicular grade I, II, III recurrent Follicle centre lymphoma, follicular grade I, II, III refractory Follicle centre lymphoma, follicular grade I, II, III stage I Follicle centre lymphoma, follicular grade I, II, III stage II Follicle centre lymphoma, follicular grade I, II, III stage III Follicle centre lymphoma, follicular grade I, II, III stage IV Follicular dendritic cell sarcoma Follicular thyroid cancer Free prostate-specific antigen increased Free prostate-specific antigen positive Fungating wound Gallbladder adenocarcinoma Gallbladder adenosquamous carcinoma Gallbladder cancer Gallbladder cancer metastatic Gallbladder cancer recurrent Gallbladder cancer stage 0 Gallbladder cancer stage I Gallbladder cancer stage II Gallbladder cancer stage III Gallbladder cancer stage IV Gallbladder neoplasm Gallbladder squamous cell carcinoma Gamma interferon therapy Gamma radiation therapy Gamma radiation therapy to bladder Gamma radiation therapy to blood Gamma radiation therapy to bone Gamma radiation therapy to brain Gamma radiation therapy to breast Gamma radiation therapy to colon Gamma radiation therapy to ear, nose, or throat Gamma radiation therapy to liver Gamma radiation therapy to lung Gamma radiation therapy to pancreas

Gamma radiation therapy to pleura

Non-Hodgkin's lymphoma unspecified histology aggressive refractory Non-Hodgkin's lymphoma unspecified histology aggressive stage I Non-Hodgkin's lymphoma unspecified histology aggressive stage II Non-Hodgkin's lymphoma unspecified histology aggressive stage III Non-Hodgkin's lymphoma unspecified histology aggressive stage IV Non-Hodgkin's lymphoma unspecified histology indolent Non-Hodgkin's lymphoma unspecified histology indolent stage I Non-Hodgkin's lymphoma unspecified histology indolent stage II Non-Hodgkin's lymphoma unspecified histology indolent stage III Non-Hodgkin's lymphoma unspecified histology indolent stage IV Nonkeratinising carcinoma of nasopharynx Non-renal cell carcinoma of kidney Non-secretory adenoma of pituitary Non-small cell lung cancer Non-small cell lung cancer metastatic Non-small cell lung cancer recurrent Non-small cell lung cancer stage 0 Non-small cell lung cancer stage I Non-small cell lung cancer stage II Non-small cell lung cancer stage III Non-small cell lung cancer stage IIIA Non-small cell lung cancer stage IIIB Non-small cell lung cancer stage IV NUT midline carcinoma Ocular cancer metastatic Ocular haemangiopericytoma Ocular lymphoma Ocular neoplasm Oesophageal adenocarcinoma Oesophageal adenocarcinoma recurrent Oesophageal adenocarcinoma stage 0 Oesophageal adenocarcinoma stage I Oesophageal adenocarcinoma stage II Oesophageal adenocarcinoma stage III Oesophageal adenocarcinoma stage IV Oesophageal cancer metastatic Oesophageal carcinoma Oesophageal carcinoma recurrent Oesophageal carcinoma stage 0 Oesophageal neoplasm Oesophageal prosthesis insertion Oesophageal squamous cell carcinoma Oesophageal squamous cell carcinoma

Undifferentiated nasopharyngeal carcinoma Undifferentiated sarcoma Ureteral neoplasm Ureteric cancer Ureteric cancer local Ureteric cancer metastatic Ureteric cancer recurrent Ureteric cancer regional Urethral cancer Urethral cancer metastatic Urethral cancer recurrent Urethral melanoma metastatic Urethral neoplasm Urethrectomy Urinary bladder sarcoma Urinary cystectomy Urinary tract carcinoma in situ Urinary tract neoplasm Uterine cancer Uterine carcinoma in situ Uterine leiomyosarcoma Uterine neoplasm Uterine tumour excision Uvulectomy Vaginal adenocarcinoma Vaginal cancer Vaginal cancer metastatic Vaginal cancer recurrent Vaginal cancer stage 0 Vaginal cancer stage I Vaginal cancer stage II Vaginal cancer stage III Vaginal cancer stage IVA Vaginal cancer stage IVB Vaginal neoplasm Vaginectomy Vascular neoplasm Vipoma Vocal cord neoplasm Vocal cordectomy Vulval cancer Vulval cancer metastatic Vulval cancer recurrent Vulval cancer stage 0 Vulval cancer stage I Vulval cancer stage II Vulval cancer stage III Vulval cancer stage IV Vulval neoplasm Vulvar adenocarcinoma Vulvectomy Waldenstrom's macroglobulinaemia Waldenstrom's macroglobulinaemia recurrent

Waldenstrom's macroglobulinaemia

metastatic

## MedDRA v20.1 Preferred Term (PT)

Gamma radiation therapy to prostate Gamma radiation therapy to skin Gamma radiation therapy to soft tissue Gamma radiation therapy to thyroid Gamma radiation therapy to uterus Gammopathy Ganglioglioma Ganglioneuroblastoma Garcin syndrome Gastrectomy Gastric cancer Gastric cancer recurrent Gastric cancer stage 0 Gastric cancer stage I Gastric cancer stage II Gastric cancer stage III Gastric cancer stage IV Gastric neoplasm Gastric sarcoma Gastric stent insertion Gastrinoma Gastrinoma malignant Gastroenteropancreatic neuroendocrine

Gastroenteropancreatic neuroendocrif tumour disease Gastrointestinal cancer metastatic Gastrointestinal carcinoma Gastrointestinal carcinoma in situ

Gastrointestinal carcinoma in situ
Gastrointestinal lymphoma
Gastrointestinal melanoma
Gastrointestinal neoplasm
Gastrointestinal stromal cancer
Gastrointestinal stromal tumour
Gastrointestinal submucosal tumour
Gastrooesophageal cancer
Genital cancer male
Genital cancer male in situ
Genital neoplasm malignant female

Genitourinary melanoma Genitourinary tract neoplasm Germ cell cancer

Germ cell cancer metastatic Germ cell neoplasm Oesophageal squamous cell carcinoma recurrent

Oesophageal squamous cell carcinoma stage 0

Oesophageal squamous cell carcinoma stage I

Oesophageal squamous cell carcinoma stage II

Oesophageal squamous cell carcinoma stage III

Oesophageal squamous cell carcinoma stage IV

Oesophagectomy Oesophagogastrectomy

Oestrogen receptor assay positive Oestrogen receptor positive breast

cancer

Oligoastrocytoma Oligodendroglioma Omentectomy

Oncogenic osteomalacia Oncologic complication Oophorectomy

Oophorectomy bilateral

Optic glioma

Optic nerve neoplasm Oral cavity cancer metastatic

Oral cavity neoplasm surgery

Oral neoplasm Orchidectomy Orchidotomy Oropharyngeal cancer

Oropharyngeal cancer recurrent

Oropharyngeal cancer stage 0 Oropharyngeal cancer stage I Oropharyngeal cancer stage II Oropharyngeal cancer stage III Oropharyngeal cancer stage IV

Oropharyngeal lymphoepithelioma Oropharyngeal neoplasm Oropharyngeal squamous cell carcinoma refractory

Waldenstrom's macroglobulinaemia stage I

Waldenstrom's macroglobulinaemia stage II

Waldenstrom's macroglobulinaemia stage III

Waldenstrom's macroglobulinaemia

stage IV

X-ray therapy to bladder X-ray therapy to blood X-ray therapy to bone X-ray therapy to brain X-ray therapy to breast X-ray therapy to colon

X-ray therapy to ear, nose, or throat

X-ray therapy to joint
X-ray therapy to liver
X-ray therapy to lung
X-ray therapy to pancreas
X-ray therapy to pleura
X-ray therapy to prostate
X-ray therapy to skin
X-ray therapy to soft tissue

X-ray therapy to thyroid X-ray therapy to uterus

X-ray treatment

Yolk sac tumour site unspecified

| SMQ PTs taken from Pseudomembranous colitis (SMQ) narrow |
|----------------------------------------------------------|

# MedDRA v20.1 Preferred Term (PT)

Clostridial infection Clostridial sepsis Clostridium bacteraemia Clostridium colitis
Clostridium difficile colitis
Clostridium difficile infection

Clostridium test positive Gastroenteritis clostridial Pseudomembranous colitis